CLINICAL TRIAL: NCT02513394
Title: PALbociclib CoLlaborative Adjuvant Study: A Randomized Phase III Trial of Palbociclib With Standard Adjuvant Endocrine Therapy Versus Standard Adjuvant Endocrine Therapy Alone for Hormone Receptor Positive (HR+) / Human Epidermal Growth Factor Receptor 2 (HER2)-Negative Early Breast Cancer
Brief Title: PALbociclib CoLlaborative Adjuvant Study
Acronym: PALLAS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance Foundation Trials, LLC. (Other)
Collaborators: Austrian Breast & Colorectal Cancer Study Group (Network); NSABP Foundation Inc (Network); PrECOG, LLC. (Other); Breast International Group (Other); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFT-05; ABCSG 42 (Other: ABCSG GmbH); BIG 14-03 (Other: Breast International Group); 2014-005181-30 (EudraCT Number)
Record Dates: First submitted 2015-07-29; First posted 2015-07-31 (Estimated); Results first posted 2022-04-13 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer
Keywords: HR+/HER2- breast cancer; Palbociclib
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): Palbociclib at a dose of 125 mg orally once daily, Day 1 to Day 21 followed by 7 days off treatment in a 28-day cycle for a total duration of 2 years, in addition to standard adjuvant endocrine therapy for a duration of at least 5 years.
  Interventions: Drug: Palbociclib; Drug: Standard Adjuvant Endocrine Therapy
- Arm B (Other): Standard adjuvant endocrine therapy for a duration of at least 5 years.
  Interventions: Drug: Standard Adjuvant Endocrine Therapy

INTERVENTIONS:
Drug: Palbociclib
  Arms: Arm A
Drug: Standard Adjuvant Endocrine Therapy

SUMMARY:
This is a prospective, two arm, international, multicenter, randomized, open-label Phase III study evaluating the addition of 2 years of palbociclib to standard adjuvant endocrine therapy for patients with HR+ / HER2- early breast cancer (EBC).

The purpose of the PALLAS study is to determine whether the addition of palbociclib to adjuvant endocrine therapy will improve outcomes over endocrine therapy alone for HR+/HER2- early breast cancer. Assessment of a variety of correlative analysis, including evaluation of the effect of palbociclib in genomically defined tumor subgroups, is planned.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to study specific procedures.
* Age ≥18 years (or per national guidelines).
* Pre- and postmenopausal women or men with Stage II (Stage IIA limited to max. 1000 patients) or Stage III early invasive breast cancer
* Patients with multicentric and/or multifocal and/or bilateral early invasive breast cancer are eligible if all histopathologically examined tumors meet pathologic criteria for ER+ and/or PR+ and HER2-.
* Patients must have histologically confirmed ER+ and/or PR+, HER2-, early invasive breast cancer.
* Patients must have undergone adequate (definitive) breast surgery for the current malignancy.

FFPE tumor tissue block must be confirmed to be received at the central sample repository prior to randomization.

* ECOG performance status 0-1.
* Patients must be able and willing to swallow and retain oral medication.
* Serum or urine pregnancy test must be negative in premenopausal women within 14 days of randomization, or in women with amenorrhea of less than 12 months at time of randomization.
* Patients who received neo/adjuvant therapy must be after last dose of chemotherapy and/or biologic therapy and must have sufficient resolution of side effects.
* Patients who received breast/axilla/post-mastectomy chest wall radiotherapy must be after last dose of radiotherapy and must have sufficient resolution of side effects.
* Patients must have sufficient resolution of any surgical side effects (no active wound healing complications).

-Patients must either be initiating or have already started adjuvant hormonal treatment. -

* Patients who already received neo/adjuvant endocrine therapy are eligible as long as they are enrolled within 12 months of initial histological diagnosis and after completing no more than 6 months of adjuvant endocrine therapy.
* Absolute neutrophil count ≥ 1,500/µL
* Platelets ≥ 100,000/ mm3
* Hemoglobin ≥ 10g/dL
* Total serum bilirubin ≤ ULN; or total bilirubin ≤ 3.0 × ULN with direct bilirubin within normal range in patients with documented Gilbert's Syndrome.
* Aspartate amino transferase (AST or SGOT) and alanine amino transferase (ALT or SGPT) ≤ 1.5 × institutional ULN.
* Serum creatinine below the upper limit of the institutional normal range (ULN) or creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with serum creatinine levels above institutional ULN.

Exclusion Criteria:

* Concurrent therapy with other Investigational Products.
* Prior therapy with any CDK inhibitor.
* Patients with Stage I or IV breast cancer are not eligible.
* History of allergic reactions attributed to compounds of chemical or biologic composition similar to palbociclib.
* Patients receiving any medications or substances that are potent inhibitors or inducers of
* CYP3A isoenzymes within 7 days of randomization.
* Uncontrolled intercurrent illness that would limit compliance with study requirements.
* Pregnant women, or women of childbearing potential without a negative pregnancy test within 14 days prior to randomization.
* Patients with a history of any malignancy are ineligible
* Patients who previously received endocrine therapy within 5 years prior to diagnosis of the current malignancy.
* Patients on antiretroviral therapy.
* Patients with clinically significant history of any chronic liver disease.
* Patients receiving concurrent exogenous hormone therapy (topical vaginal estrogen therapy is allowable).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5796 (Actual)
Dates: Start 2015-08; Primary Completion 2020-11 (Actual); Study Completion 2028-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Evanthia Galanis, MD, Principal Investigator — Alliance Foundation Trials, LLC.; Erica Mayer, MD, Principal Investigator — Dana-Farber Cancer Institute; Angela DeMichele, MD, Principal Investigator — University of Pennsylvania; Michael Gnant, MD, Principal Investigator — ABCSG, Medical University Vienna
Locations (437):
- United States (192):
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Southern Cancer Center PC - Providence, Mobile, Alabama
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Cancer Center, Anchorage, Alaska
  - Mayo Clinic in Arizona, Phoenix, Arizona
  - Kaiser Permanente Anaheim Medical Center, Anaheim, California
  - Kaiser Permanente Baldwin Park Medical Center, Baldwin Park, California
  - Kaiser Permanente Bellflower Medical Center, Bellflower, California
  - Kaiser Permanente Fontana Medical Center, Fontana, California
  - Marin Cancer Care, Greenbrae, California
  - Marin Cancer Center, Greenbrae, California
  - Kaiser Permanente Harbor City Medical Center, Harbor City, California
  - Kaiser Permanente Irvine Medical Center, Irvine, California
  - UCSD Moores Cancer Center, La Jolla, California
  - Long Beach Memorial Medical Center - Todd Cancer Institute, Long Beach, California
  - Kaiser Permanente Sunset Medical Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Kaiser Permanente Oakland Medical Center, Oakland, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Kaiser Permanente Panorama City Medical Center, Panorama City, California
  - Kaiser Permanente Riverside Medical Center, Riverside, California
  - Kaiser Permanente Roseville Medical Center, Roseville, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - University of California, San Diego, California
  - Kaiser Permanente San Diego Medical Center, San Diego, California
  - Sharp Memorial Hospital, San Diego, California
  - Kaiser Permanente San Francisco Medical Center, San Francisco, California
  - UCSF Helen Diller Comprehensive Cancer Center, San Francisco, California
  - Kaiser Permanente San Jose Medical Center, San Jose, California
  - Kaiser Permanente San Leandro Medical Center, San Leandro, California
  - Kaiser Permanente San Marcos Medical Center, San Marcos, California
  - Kaiser Permanente Santa Clara Medical Center, Santa Clara, California
  - Kaiser Permanente South San Francisco Medical Center, South San Francisco, California
  - Stanford Women's Cancer Center, Stanford, California
  - Kaiser Permanente Vallejo Medical Center, Vallejo, California
  - Kaiser Permanente Walnut Creek Medical Center, Walnut Creek, California
  - Kaiser Permanente Cadillac Medical Center, West Los Angeles, California
  - Kaiser Permanente Woodland Hills Medical Center, Woodland Hills, California
  - Western States Cancer Research NCORP, Denver, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Memorial Sloan Cancer Center - Hartford Healthcare Center Institute at HOCC, New Britain, Connecticut
  - Christiana Health System - Christiana Hospital, Newark, Delaware
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - George Washington University Medical Faculty Associates, Washington D.C., District of Columbia
  - Morton Plant Hospital, Clearwater, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Miami Miller School of Medicine Sylvester Cancer Center, Miami, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Advent Health Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Cancer Center LAPS, Chicago, Illinois
  - Cancer Care Specialist of Central Illinois, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - NorthShore University Health System - Evanston Hospital, Evanston, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Joliet Oncology Hematology Associates Limited, Joliet, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Anthony Medical Center, Rockford, Illinois
  - Orchard Healthcare Research Inc., Skokie, Illinois
  - NorthShore Hematology Oncology-Libertyville, Skokie, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Indiana University - Melvin and Bren Simon Cancer Center LAPS, Indianapolis, Indiana
  - IU Health Ball Memorial Hospital, Muncie, Indiana
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - McFarland Clinic, P.C., Ames, Iowa
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Iowa Oncology Research Assoc, Des Moines, Iowa
  - Medical Oncology and Hematology Associates - Des Moines, Des Moines, Iowa
  - Covenant Medical Center, Waterloo, Iowa
  - University of Kentucky-Markey Cancer Center, Lexington, Kentucky
  - Norton Cancer Institute - Brownsboro, Louisville, Kentucky
  - Ochsner Medical Center, New Orleans, Louisiana
  - Eastern Maine Medical Center d/b/a Northern Light Cancer Institute, Bangor, Maine
  - New England Cancer Specialists - Scarborough, Scarborough, Maine
  - Anne Arundel Medical Center, Annapolis, Maryland
  - Mercy Medical Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - MedStar Good Samaritan Hospital, Baltimore, Maryland
  - MedStar Franklin Square Medical Center Winberg Cancer Institute, Baltimore, Maryland
  - Medstar Union Memorial Hospital, Baltimore, Maryland
  - JHU Sidney Kimmel Comprehensive Cancer Center LAPS, Baltimore, Maryland
  - Frederick Regional Health System James M Stockman Cancer Institute, Baltimore, Maryland
  - Maryland Oncology Hematology PA, Bethesda, Maryland
  - Tidal Health Peninsula Regional, Salisbury, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Beth Israel Deaconess Hospital - Plymouth Jordan Club Cancer Center, Plymouth, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Spectrum Health Butterworth Research Pharmacy, Grand Rapids, Michigan
  - Trinity Health Michigan, Livonia, Michigan
  - Essentia Health NCORP, Duluth, Minnesota
  - Mayo Clinic-Rochester, Rochester, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Metro Minnesota Oncology Research Consortium, Saint Louis Park, Minnesota
  - St. Luke's Hospital, Kansas City, Missouri
  - Phelps Country Regional Medical Center, Rolla, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Nebraska Hematology and Oncology, Lincoln, Nebraska
  - Southeast Nebraska Cancer Center, Lincoln, Nebraska
  - Cancer Alliance of Nebraska, Omaha, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - New Hampshire Oncology-Hematology PA, Concord, Concord, New Hampshire
  - New Hampshire Oncology-Hematology PA, Hooksett, New Hampshire
  - Solinsky Center for Cancer Care, Hooksett, New Hampshire
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Norris Cotton Cancer Center - Nashua, Lebanon, New Hampshire
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Rutgers Cancer Center Institute of New Jersey, New Brunswick, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Hematology Oncology Associates of Central New York - East Syracuse, East Syracuse, New York
  - Queens Hospital Center, Jamaica, New York
  - Northwell Health NCORP, New Hyde Park, New York
  - Beth Israel Medical Center - New York, New York, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Memorial Sloan Kettering Cancer Center - LAPS, New York, New York
  - Oneonta FoxCare Center, Oneonta, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Einstein Campus, The Bronx, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - The Charlotte-Mecklenburg Hospital Authority, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Kinston Medical Specialists, PA, Kinston, North Carolina
  - First Health of the Carolinas - Moore Regional Hospital, Pinehurst, North Carolina
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Cleveland Clinic Cancer Center/Hillcrest Hospital, Mayfield Heights, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Providence Portland Medical Center, Portland, Oregon
  - Hematology & Oncology Associates of Northeastern PA, Dunmore, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Hospital of the University of Pennsylvania Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC MaGee Women's Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute- Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Reading Hospital/McGlinn Cancer Institute, Wyomissing, Pennsylvania
  - WellSpan Health York Cancer Center, York, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - Lexington Medical Center/Lexington Oncology Associates, Columbia, South Carolina
  - Avera Cancer Institute-Aberdeen, Aberdeen, South Dakota
  - Monument Health Rapid City Hospital, Rapid City, South Dakota
  - Rapid City Regional Hospital/Regional Cancer Care Institute, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Nashville General Hospital at Meharry, Nashville, Tennessee
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Houston Methodist Hospital Cancer Center, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Doctors Hospital of Laredo, Laredo, Texas
  - Huntsman Cancer Institute - University of Utah, Salt Lake City, Utah
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - VCU Massey Cancer Center, Richmond, Virginia
  - CAMC Cancer Center, Charleston, West Virginia
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - HSHS Saint Vincent Hospital, Green Bay, Wisconsin
  - Gunderson Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Wheaton Franciscan Healthcare - St. Joseph, Milwaukee, Wisconsin
  - Columbia St. Mary's Water Tower Medical Commons, Milwaukee, Wisconsin
  - Wheaton Franciscan Healthcare-All Saints, Racine, Wisconsin
  - Orchard Healthcare Research Inc., Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Wheaton Franciscan Healthcare - Wauwatosa, Wauwatosa, Wisconsin
- Australia (21):
  - Southern Highlands Cancer Centre, Bowral, New South Wales
  - Coffs Harbour Health Campus - MNCCI, Coffs Harbour, New South Wales
  - The Breast & Endocrine Centre, Gateshead, New South Wales
  - Gosford Hospital, Gosford, New South Wales
  - Macquarie University Hospital, Macquarie Park, New South Wales
  - Orange Health Service, Orange, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Royal Brisbane & Women's Hospital, Brisbane, Queensland
  - Flinders Drive, Bedford Park, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - The Northern Hospital, Epping, Victoria
  - St Vincent's Hospital, Fitzroy, Victoria
  - Peninsula Health - Frankston Hospital, Frankston, Victoria
  - University Hospital, Geelong, Geelong, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Peninsula Health - Frankston Hospital, Melbourne, Victoria
  - Western Health, Sunshine Hospital, St Albans, Victoria
  - South West Healthcare, Warrnambool, Warrnambool, Victoria
  - St John of God Bunbury Hospital, Bunbury, Western Australia
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Breast Cancer Research Centre - WA, Nedlands, Western Australia
- Austria (24):
  - LKH Feldkirch, Department of Internal Medicine, Feldkirch
  - LKH Univ Klinikum Graz, Dept of Internal Med. and Oncology, Graz
  - Medical University of Graz, Gyn. Dept., Graz
  - University Hospital Innsbruck, Department of Obstetrics and Gynaecology, Innsbruck
  - BKH Kufstein, Innere Medizin, Kufstein
  - LKH Hochsteiermark Leoben, Leoben
  - Hospital of the Sisters of Charity Linz, Surg. Dept., Breast Health Center, Linz
  - Kepler Universitätsklinikum Med. Campus III, Linz
  - Weinviertelklinikum Mistelbach, Department of Surgery, Mistelbach
  - BHS Ried, Abt. f. Gynäkologie, Ried
  - LKH Salzburg, Univ. Klinik f. Innere Med. III, Salzburg
  - Universitätsklinikum St. Pölten, Innere Medizin, Sankt Pölten
  - Breast Centre Dr. Wette Viktor, Sankt Veit an der Glan
  - Phyrn-Eisenwurzen Klinikum Steyr, Steyr
  - Medical University of Vienna Department of Obstetrics and Gynaecology, Vienna
  - Medical University Vienna - Coop Group Surgery/Oncology, Vienna
  - Hospital Hietzing, Gynecology, Vienna
  - St. Josef Krankenhaus, Department of Internal I, Vienna
  - Klinik Ottakring, Vienna
  - Salzkammergut-Klinikum Vöcklabruck, Vöcklabruck
  - Brustordination Dr. Thiel, Weiz
  - Klinikum Wels - Grieskirchen GmbH, Department of Internal Medicine IV, Wels
  - Landesklinikum Wr. Neustadt, Department of Surgery, Wiener Neustadt
  - LKH Wolfsberg, Department of Surgery, Wolfsberg
- Belgium (12):
  - OLV ziekenhuis Aalst/Radiotherapy-Oncology, Aalst
  - CHU Saint Pierre/Medical Oncology, Brussels
  - Institut Jules Bordet/Medical Oncology Department, Brussels
  - Cliniques Universitaires Saint-Luc, Oncologisch centrum, Brussels
  - Grand Hopital de Charleroi - Oncologie-hématologie, Charleroi
  - University Hospital Antwerp (UZA), Edegem
  - UZ Leuven/ Gynaecologie-Oncologie, Leuven
  - CHC - Saint-Joseph/Oncology-Hematology, Liège
  - CHU Sart Tilman Liège (Medical Oncology), Liège
  - Clinique et Maternite Sainte-Elisabeth - Oncology Department, Namur
  - CHR - Centre Hospitalier Peltzer La Tourelle/ Oncology Department, Verviers
  - GZA Ziekenhuizen (Campus Sint-Augustinus) / Oncologische Centrum, Wilrijk
- Canada (19):
  - Tom Baker Cancer Centre - Dept. of Oncology, Calgary, Alberta
  - BC Cancer Agency- Abbotsford Centre, Abbotsford, British Columbia
  - BC Cancer Agency - Sindi Ahluwalia Hawkins Centre for the Southern Interior, Kelowna, British Columbia
  - BC Cancer Agency - Vancouver Cancer Centre, Vancouver, British Columbia
  - CancerCare Manitoba - St. Boniface Hospital, Winnipeg, Manitoba
  - The Vitalite Health Network - Dr. Leon Richard, Moncton, New Brunswick
  - Horizon Health Network - Saint John Regional Hospital, Saint John, New Brunswick
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Kingston General Hospital, Cancer Centre of Southeastern Ontario/Oncology, Kingston, Ontario
  - Grand River Regional Cancer Center, Kitchener, Ontario
  - Niagara Health System, St. Catharines, Ontario
  - Sunnybrook, Toronto, Ontario
  - University Health Network Princess Margaret Cancer Centre, Toronto, Ontario
  - The Jewish General Hospital, Montreal, Quebec
  - CHUM Hôtel Dieu, Montreal, Quebec
  - CHU de Québec - Hôpital du St Sacrement, Québec, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Center, University of Saskatchewan, Saskatoon, Saskatchewan
- Germany (27):
  - University Hospital Aachen, Aachen
  - Praxisklinik Krebsheilkunde für Frauen, Berlin
  - Helios Klinikum Berlin-Buch, Berlin
  - Studienzentrum City, Berlin
  - Marienhospital Bottrop, Klinik für Gynäkologie und Geburtshilfe, Bottrop
  - Studien GbR Braunschweig, Lorenz&HeckerWesche, Braunschweig
  - Praxis und Tagesklinik für gynäkologische Onkologie,, Ebersberg
  - MVZ Eggenfelden, Eggenfelden
  - Frauenklinik/University Hospital Erlangen, Erlangen
  - Centrum für Hämatologie und Onkologie Bethanien, Frankfurt
  - Agaplesion Markus Krankenhaus, Frankfurt
  - Klinikum Frankfurt Höchst, Frankfurt
  - Onkol. GP Dres. med. Wilke/Wagner/Petzoldt, Fürth
  - Universitätsfrauenklinik Halle (Saale), Halle
  - University Medical Center Hamburg-Eppendorf, Department of Gynecology, Hamburg
  - Albertinen Krankenhaus, Hamburg
  - Städtisches Klinikum Karlsruhe, Karlsruhe
  - Elisabeth Krankenhaus Kassel Brustzentrum, Kassel
  - St. Elisabeth Krankenhaus Leipzig, Leipzig
  - St. Vincenz KH Limburg Frauenklinik, Limburg
  - UKSH Campus Lübeck, Klinik für Frauenheilkunde und Geburtshilfe, Lübeck
  - Universitätsmedizin Mainz, Mainz
  - Praxis Gynäkologie Arabella, München
  - University Clinic Oldenburg, Oldenburg
  - Oncologianova GmbH, Recklinghausen
  - HELIOS Klinik Rottweil - Gynäkologie, Rottweil
  - St. Josefs-Hospital, Wiesbaden
- Hungary (5):
  - Országos Onkológiai Intézet - "B" Belgyógyászati Onkológiai és Klinikai Farmakológiai Osztály, Budapest
  - Uzsoki Utcai Kórház - Onkoradiológia, Sugárterápia, Fővárosi Onkoradiológiai Központ, Budapest
  - University of Debrecen Medical Center, Clinic of Oncology, Debrecen
  - Petz Aladár Megyei Oktatókórház - Onkoradiológiai Osztály, Győr
  - Szegedi Tudomanyegyetem Általános Orvostudományi Kar Szent-Györgyi Albert Klinikai Központ, Onkoterápiás Klinika, Szeged
- Ireland (9):
  - Bon Secours Hospital, Cork, Cork
  - Cork University Hospital, Oncology Clinical Trials Unit, Cork
  - Beaumont Hospital - Cancer Clinical Trials Unit, Dublin
  - Mater Misericordiae University Hospital, Dublin
  - St James's Hospital, Cancer Clinical Trials Office, Old Admin Building,, Dublin
  - St Vincent Hospital - Medical Oncology Research Department, Dublin
  - University Hospital Limerick, Midwestern Cancer Centre, Limerick
  - Sligo University Hospital, Sligo
  - University Hospital Waterford, Cancer Research Department, Waterford
- Israel (3):
  - Rabin Medical Center (RMC), Petah Tikva, Central District
  - Sheba Medical Center Tel Hashomer, Ramat Gan, Tel Aviv
  - Sourasky Medical Center, Tel Aviv
- Italy (13):
  - Azienda Ospedaliero-Universitaria di Ferrara, Ferrara
  - Azienda Ospedaliero-Universitaria Careggi/Florence University/Radiation Oncology Unit, Florence
  - Department of Internal Medicine (DIMI) - IRCCS San Martino University Hospital, Genoa
  - P.O. Misericordia AUSL Toscana Sud Est, Grosseto
  - Ospedale "Mater Salutis" di Legnago, Dept. of Medical Oncology, Legnago
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (I.R.S.T.) IRCCS, Meldola
  - Ospedale San Raffaele, Milan
  - Istituto Europeo di Oncologia, Milan
  - Policlinico di Monza - Istituto di Oncologia del Policlinico di Monza, Monza
  - Medical Oncology Unit; University Hospital of Parma (Azienda Ospedaliero-Universitaria di Parma), Parma
  - Nuovo Ospedale di Prato (NOP) - Azienda USL4 Prato, Prato
  - ASST Bergamo Ovest, Treviglio
  - S. Anna Hospital (Ospedale Sant'Anna)- Turin, Turin
- Japan (6):
  - Nagoya City University Hospital/Dept. of Breast & Endocrine Surgery, Nagoya, Aichi-ken
  - Department of Breast Surgery National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Chiba Cancer Center, Chiba
  - Kyoto University Hospital/Breast Surgery, Kyoto
  - National Hospital Organization Osaka National Hospital, Osaka
  - Osaka International Cancer Institute, Osaka
- Mexico (3):
  - Centro Médico Zambrano Hellion, Monterrey, Nuevo León
  - Centro Oncológico Estatal ISSEMYM, Toluca, Toluca
  - National Cancer Institute Mexico, Breast Cancer Department, Mexico City
- Netherlands (6):
  - Máxima Medisch Centrum, Eindhoven
  - Zuyderland Ziekenhuis, Oncology, Geleen
  - St Antonius Hospital, Nieuwegein
  - Hagaziekenhuis, The Hague
  - Zaans Medical Center, Zaandam
  - Isala, Dept of Medical Oncology, Zwolle
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne (UCK), Klinika Onkologii I Radioterapii, Gdansk
  - Instytut MSF Spółka z ograniczoną odpowiedzialnością, Lodz
  - Opolskie Centrum Onkologii, Oddzial Onkologii Klinicznej, Opole
  - Klinika Nowotworów Piersi i Chirurgii Rekonstrukcyjnej, Centrum Onkologii-Instytut im. Marii Skłodowskiej-Curie, Warsaw
- Portugal (5):
  - Instituto Português de Oncologia (IPO) de Lisboa Francisco Gentil, Lisbon
  - Centro Clinico Champalimaud, Lisbon
  - Hospital da Luz, Lisbon
  - CUF Descobertas Hospital, Hemato-Oncologia, Lisbon
  - Instituto Português de Oncologia (IPO) Francisco Gentil do Porto, Porto
- South Korea (3):
  - Seoul National University Hospital, Hematology-Medical Oncology, Seoul
  - Severance Hospital Medical Doctor at Department of Medical Oncology, Seoul
  - Samsung Medical Centre, Breast Cancer Center, Department of Medicine, Division of Hematology/Oncology, Seoul
- Spain (46):
  - Complejo Hospitalario Universitario A Coruña (CHUAC), A Coruña
  - Centro Oncologico de Galicia, A Coruña
  - Hospital General Universitario Alicante, Alicante
  - ICO Badalona, Badalona
  - Hospital del Mar, Barcelona
  - Hospital Universitari Quirón Dexeus, Barcelona
  - Hospital Clinic Barcelona, Barcelona
  - Hospital General de Granollers, Barcelona
  - Instituto Catalán de Oncología (ICO) de L'Hospitalet de Llobregat, Barcelona
  - Hospital Vall d´Hebron, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Consorcio Hospitalario Provincial de Castellon, Castellon
  - San Pedro de Alcántara, Cáceres
  - Hospital Reina Sofía, Córdoba
  - Hospital General Universitario de Elche, Elche
  - ICO/ H. Josep Trueta, Girona
  - Complejo asistencial universitario de Leon, León
  - Hospital Universitario Gregorio Marañón, Madrid
  - MD Anderson Cancer Center, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital La Paz, Servicio de Oncologia Médica, Madrid
  - CIOCC - Centro Integral Oncológico Clara Campal / Hospital HM Universitario Sanchinarro, Madrid
  - Hospital Puerta de Hierro Majadahonda, Oncologia Médica, Madrid
  - Hospital Universitario Fundacion Alcorcón, Madrid
  - Hospital Clínico Universitario Virgen de la Victoria, Málaga
  - Hospital General Universitario José Mª Morales Meseguer, Murcia
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospitali Universitari son Espases, Palma
  - Hospital Son Llatzer, Palma
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Universitari Sant Joan de Reus, Reus
  - Hospital Universitario Donostia, San Sebastián
  - Hospital de Sant Juan Despi Moisés Broggi, Sant Joan Despì
  - Hospital Clinico Universitario de Santiago, Santiago
  - Hospital Unversitario Virgen Macarena, Seville
  - Hospital Quirón Sagrado Corazón, Seville
  - Hospital Universitario Virgen del Rocio, Seville
  - Consorci Sanitari de Terrassa, Terrassa
  - Hospital Virgen de la Salud, Toledo
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hosital Arnau de Vilanova Valencia, Valencia
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza
- Sweden (5):
  - Gävle Hospital, Dept. of Oncology, Gävle
  - Sahlgrenska University Hospital, Dept. Oncology, Gothenburg
  - Universitetssjukhuset Örebro (University Hospital) Örebro, Onkologkliniken, Örebro
  - Karolinska Universitetssjukhuset, Bröstcentrum A2:00, Stockholm
  - Akademiska Sjukhuset Uppsala (University Hospital), Onkologkliniken, Uppsala
- Switzerland (13):
  - Kantonspital Baden, Baden, Canton of Aargau
  - Spital STS AG, Onkologiezentrum Thun-Berner Oberland, Thun, Canton of Bern
  - Hôpitaux Universitaires de Genève, Geneva, Canton of Geneva
  - IOSI-Breast Cancer Unit-Ospedale San Giovanni-Bellinzona, Bellinzona, Canton Ticino
  - Fondazione Oncologia Lago Maggiore, Locarno, Locarno, Canton Ticino
  - Kantonsspital Graubünden, Chur, Kanton Graubünden
  - Dep. Oncology, University Hospital, Basel
  - HFR Fribourg, Oncology Department, Fribourg
  - Luzerner Kantonsspital, Dept. of Medical Oncology, Lucerne
  - Onkologisches Forschungszentrum Klinik St. Anna, Hirslanden, Lucerne
  - Kantonsspital St.Gallen, Onkologie/Hämatologie, Sankt Gallen
  - Brust-Zentrum Zürich, Zurich
  - Universitätsspital Zürich, Klinik für Onkologie, Zurich
- Taiwan (5):
  - Changhua Christian Hospital/General Surgery, Changhua, Changhua County
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Division of Hemato-Oncology, Dept. Internal Medicine, Tainan
  - National Taiwan University Hospital/Department of Surgery, Taipei
  - Taipei Veterans General Hospital/General Surgery, Taipei
- United Kingdom (16):
  - City Hospital Birmingham, Birmingham
  - University Hospitals Bristol NHS Foundation Trust, Bristol
  - Velindre Cancer Centre, Cardiff
  - Royal Marsden Hospital Chelsea, Chelsea
  - The Beatson West of Scotland Cancer Centre, Glasgow
  - University Hospitals of Leicester, Leicester
  - Royal Liverpool University Hospital, Liverpool
  - Guy's and St Thomas' NHS Foundation Trust, London
  - The Royal Marsden Sutton, London
  - Charing Cross Hospital, London
  - Maidstone Hospital, Kent Oncology Centre, Maidstone
  - The Christie NHS Foundation Trust, Manchester
  - Northern Centre for Cancer Care, Newcastle upon Tyne
  - Nottingham University Hospitals NHS TRUST UK, Nottingham
  - Weston Park Hospital, Sheffield Teaching Hospitals, Sheffield
  - Royal Cornwall Hospitals NHS Trust, Oncology Trials, Sunrise Centre, Truro

REFERENCES:
- [Derived] Shinn E, Zahrieh D, DeMichele A, Zdenkowski N, Lemieux J, Mao J, Bjelic-Radisic V, Naughton MJ, Pfeiler G, Gelmon K, Balko JM, Egle D, Zoppoli G, Traina T, Jimenez MM, Novoa SA, Haddad T, Chan A, Ring A, Wolff A, Symmans WF, Ponce Lorenzo J, Sabanathan D, Burstein HJ, Nowecki ZI, Pristauz-Telsnigg G, Brufsky A, Bellet-Ezquerra M, Foukakis T, Novik Y, Rubovszky G, Singer CF, Muehlbacher K, Filho OM, Goulioti T, Law E, Partridge AH, Carey LA, Zoroufy A, Hlauschek D, Fesl C, Mayer EL, Gnant M. Impact of adding palbociclib on treatment adherence to ongoing adjuvant endocrine treatment in the global randomized PALLAS randomized trial in patients with early breast cancer. Breast Cancer Res Treat. 2025 Jun;211(2):385-397. doi: 10.1007/s10549-025-07653-2. Epub 2025 Mar 27. PMID 40140172
- [Derived] DeMichele A, Dueck AC, Hlauschek D, Martin M, Burstein H, Pfeiler G, Zdenkowski N, Wolff A, Bellet-Ezquerra M, Winer E, Balic M, Miller K, Colleoni M, Lake D, Rubovsky G, Cameron D, Balko J, Singer CF, Nowecki Z, Iwata H, Wolmark N, Parraga KA, Rugo H, Steger GG, Traina T, Werutsky G, Czajkowska D, Metzger O, El-Abed S, Theall KP, Lu RD, O'Brien P, Fesl C, Mayer E, Gnant M. Outcomes in stage IIA versus stage IIB/III in the PALLAS trial [ABCSG-42/AFT-05/PrE0109/BIG-14-13]). Breast Cancer Res. 2025 Jan 23;27(1):12. doi: 10.1186/s13058-024-01941-3. PMID 39849600
- [Derived] Pfeiler G, Hlauschek D, Mayer EL, Deutschmann C, Kacerovsky-Strobl S, Martin M, Meisel JL, Zdenkowski N, Loibl S, Balic M, Park H, Prat A, Isaacs C, Bajetta E, Balko JM, Bellet-Ezquerra M, Bliss J, Burstein H, Cardoso F, Fohler H, Foukakis T, Gelmon KA, Goetz M, Haddad TC, Iwata H, Jassem J, Lee SC, Linderholm B, Los M, Mamounas EP, Miller KD, Morris PG, Munzone E, Gal-Yam EN, Ring A, Shepherd L, Singer C, Thomssen C, Tseng LM, Valagussa P, Winer EP, Wolff AC, Zoppoli G, Machacek-Link J, Schurmans C, Huang X, Gauthier E, Fesl C, Dueck AC, DeMichele A, Gnant M; PALLAS Groups and Investigators. Impact of BMI in Patients With Early Hormone Receptor-Positive Breast Cancer Receiving Endocrine Therapy With or Without Palbociclib in the PALLAS Trial. J Clin Oncol. 2023 Nov 20;41(33):5118-5130. doi: 10.1200/JCO.23.00126. Epub 2023 Aug 9. PMID 37556775
- [Derived] Mayer EL, Fesl C, Hlauschek D, Garcia-Estevez L, Burstein HJ, Zdenkowski N, Wette V, Miller KD, Balic M, Mayer IA, Cameron D, Winer EP, Ponce Lorenzo JJ, Lake D, Pristauz-Telsnigg G, Haddad TC, Shepherd L, Iwata H, Goetz M, Cardoso F, Traina TA, Sabanathan D, Breitenstein U, Ackerl K, Metzger Filho O, Zehetner K, Solomon K, El-Abed S, Theall KP, Lu DR, Dueck A, Gnant M, DeMichele A. Treatment Exposure and Discontinuation in the PALbociclib CoLlaborative Adjuvant Study of Palbociclib With Adjuvant Endocrine Therapy for Hormone Receptor-Positive/Human Epidermal Growth Factor Receptor 2-Negative Early Breast Cancer (PALLAS/AFT-05/ABCSG-42/BIG-14-03). J Clin Oncol. 2022 Feb 10;40(5):449-458. doi: 10.1200/JCO.21.01918. Epub 2022 Jan 7. PMID 34995105
- [Derived] Gnant M, Dueck AC, Frantal S, Martin M, Burstein HJ, Greil R, Fox P, Wolff AC, Chan A, Winer EP, Pfeiler G, Miller KD, Colleoni M, Suga JM, Rubovsky G, Bliss JM, Mayer IA, Singer CF, Nowecki Z, Hahn O, Thomson J, Wolmark N, Amillano K, Rugo HS, Steger GG, Hernando Fernandez de Aranguiz B, Haddad TC, Perello A, Bellet M, Fohler H, Metzger Filho O, Jallitsch-Halper A, Solomon K, Schurmans C, Theall KP, Lu DR, Tenner K, Fesl C, DeMichele A, Mayer EL; PALLAS groups and investigators. Adjuvant Palbociclib for Early Breast Cancer: The PALLAS Trial Results (ABCSG-42/AFT-05/BIG-14-03). J Clin Oncol. 2022 Jan 20;40(3):282-293. doi: 10.1200/JCO.21.02554. Epub 2021 Dec 7. PMID 34874182
- [Derived] Mayer EL, Dueck AC, Martin M, Rubovszky G, Burstein HJ, Bellet-Ezquerra M, Miller KD, Zdenkowski N, Winer EP, Pfeiler G, Goetz M, Ruiz-Borrego M, Anderson D, Nowecki Z, Loibl S, Moulder S, Ring A, Fitzal F, Traina T, Chan A, Rugo HS, Lemieux J, Henao F, Lyss A, Antolin Novoa S, Wolff AC, Vetter M, Egle D, Morris PG, Mamounas EP, Gil-Gil MJ, Prat A, Fohler H, Metzger Filho O, Schwarz M, DuFrane C, Fumagalli D, Theall KP, Lu DR, Bartlett CH, Koehler M, Fesl C, DeMichele A, Gnant M. Palbociclib with adjuvant endocrine therapy in early breast cancer (PALLAS): interim analysis of a multicentre, open-label, randomised, phase 3 study. Lancet Oncol. 2021 Feb;22(2):212-222. doi: 10.1016/S1470-2045(20)30642-2. Epub 2021 Jan 15. PMID 33460574
- [Derived] Dieras V, Rugo HS, Schnell P, Gelmon K, Cristofanilli M, Loi S, Colleoni M, Lu DR, Mori A, Gauthier E, Huang Bartlett C, Slamon DJ, Turner NC, Finn RS. Long-term Pooled Safety Analysis of Palbociclib in Combination With Endocrine Therapy for HR+/HER2- Advanced Breast Cancer. J Natl Cancer Inst. 2019 Apr 1;111(4):419-430. doi: 10.1093/jnci/djy109. PMID 30032196

RESULTS

PARTICIPANT FLOW:
Groups:
- Palbociclib Plus Endocrine Therapy (Arm A): Palbociclib at a dose of 125 mg orally once daily, Day 1 to Day 21 followed by 7 days off treatment in a 28-day cycle for a total duration of 2 years, in addition to standard adjuvant endocrine therapy for a duration of at least 5 years.
- Endocrine Therapy Alone (Arm B): Standard adjuvant endocrine therapy for a duration of at least 5 years.
Period: Overall Study
Arm/Group | Palbociclib Plus Endocrine Therapy (Arm A) | Endocrine Therapy Alone (Arm B)
Started | 2896 | 2900
Completed | 2884 | 2877
Not Completed | 12 | 23
Not completed — Withdrawal by Subject | 11 | 23
Not completed — Ineligible | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Palbociclib Plus Endocrine Therapy (Arm A) | Endocrine Therapy Alone (Arm B) | Total
Number analyzed (Participants) | 2884 | 2877 | 5761
Age, Continuous [Median (Full Range); unit: years] | 52 [25 to 90] | 52 [22 to 85] | 52 [22 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2867 | 2858 | 5725
  Male | 17 | 19 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 138 | 127 | 265
  Not Hispanic or Latino | 2504 | 2532 | 5036
  Unknown or Not Reported | 242 | 218 | 460
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asain | 138 | 141 | 279
  Race: Black or African American/African Heritage | 74 | 75 | 149
  Race: White | 2521 | 2498 | 5019
  Race: Native Hawaiian or other Pacific Islander | 4 | 8 | 12
  Race: American Indian or Alaska Native | 14 | 22 | 36
  Race: Other | 37 | 36 | 73
  Race: Unknown | 96 | 97 | 193

OUTCOME MEASURES:

1. Primary Outcome: Invasive Disease Free Survival (iDFS)
Description: Invasive disease-free survival (iDFS) for the combination of at least 5 years endocrine therapy and 2-year palbociclib treatment versus at least 5 years endocrine therapy alone in patients with histologically confirmed HR+/HER2- invasive early breast cancer (EBC) at 4 years. iDFS is defined as the time from randomization to the date of the first event: local/regional invasive ipsilateral recurrence, contralateral invasive breast cancer, distant recurrence, second primary invasive cancer of non-breast origin or death from any cause. Direct comparison between arms used time to iDFS events and Kaplan-Meier Log-rank analysis. Due to the medians not yet achieved, the percentage of patients considered iDFS at 4 years is reported.
Time Frame: 4 years
Measure: Number; unit: percentage of participants
Arm/Group | Palbociclib Plus Endocrine Therapy (Arm A) | Endocrine Therapy Alone (Arm B)
Number analyzed (Participants) | 2884 | 2877
percentage of participants | 84.2 | 84.5
Statistical Analysis 1: Comparison: Palbociclib Plus Endocrine Therapy (Arm A) vs Endocrine Therapy Alone (Arm B); Test type: Other; p = 0.65, Log Rank; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.81 to 1.14] — This two sided p value was stratified by (neo)adjuvant chemotherapy (yes vs no) and age (<=50 vs >50)

2. Secondary Outcome: Invasive Disease Free Survival (iDFS) Excluding Second Primary Invasive Cancers of Non-breast Origin.
Description: Invasive disease-free survival (iDFS, excluding second primary invasive cancers of non-breast origin) for the combination of at least 5 years endocrine therapy and 2-year palbociclib treatment versus at least 5 years endocrine therapy alone in patients with histologically confirmed HR+/HER2- invasive early breast cancer (EBC) at 4 years. iDFS excluding second primary invasive cancers of non-breast origin is defined as the time from randomization to the date of the first event: local/regional invasive ipsilateral recurrence, contralateral invasive breast cancer, distant recurrence, or death from any cause. Second primary invasive cancers of non-breast origin will not be considered as events for this endpoint. Direct comparison between arms used time to iDFS events and Kaplan-Meier Log-rank analysis. Due to the medians not yet achieved, the percentage of patients considered iDFS at 4 years is reported.
Time Frame: 4 years
Measure: Number; unit: percentage of patients
Arm/Group | Palbociclib Plus Endocrine Therapy (Arm A) | Endocrine Therapy Alone (Arm B)
Number analyzed (Participants) | 2884 | 2877
percentage of patients | 85.4 | 86.0
Statistical Analysis 1: Comparison: Palbociclib Plus Endocrine Therapy (Arm A) vs Endocrine Therapy Alone (Arm B); Test type: Other; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.82 to 1.19]

3. Secondary Outcome: Distant Recurrence-free Survival (DRFS)
Description: Compare time to distant recurrence-free survival (DRFS). Distant recurrence is defined according to STEEP criteria as the time from randomization to the date of the first event: distant recurrence or death from any cause. Patients with a locoregional recurrence will continue to be followed for DRFS. Surviving patients who are event-free will be censored at: the date of last disease assessment, or withdrawal of consent to be followed, or death whichever came first. Direct comparison between arms used time to DRFS events and Kaplan-Meier Log-rank analysis. Due to the medians not yet achieved, the percentage of patients considered DRFS at 4 years is reported.
Time Frame: 4 years
Measure: Number; unit: percentage of patients
Arm/Group | Palbociclib Plus Endocrine Therapy (Arm A) | Endocrine Therapy Alone (Arm B)
Number analyzed (Participants) | 2884 | 2877
percentage of patients | 86.2 | 87.8
Statistical Analysis 1: Comparison: Palbociclib Plus Endocrine Therapy (Arm A) vs Endocrine Therapy Alone (Arm B); Test type: Other; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.87 to 1.28]

4. Secondary Outcome: Overall Survival (OS)
Description: Compare overall survival (OS). Overall survival is defined as the time period between randomization and death. Surviving patients classified as lost-to-follow up or having withdrawn consent to be followed will be censored at their date of last contact or withdrawal of consent to be followed, whichever occurs first.
Time Frame: 4 years
Measure: Number; unit: percentage of patients
Arm/Group | Palbociclib Plus Endocrine Therapy (Arm A) | Endocrine Therapy Alone (Arm B)
Number analyzed (Participants) | 2884 | 2877
percentage of patients | 93.8 | 95.2
Statistical Analysis 1: Comparison: Palbociclib Plus Endocrine Therapy (Arm A) vs Endocrine Therapy Alone (Arm B); Test type: Other; Hazard Ratio (HR) = 1.32, 95% CI 2-sided [0.98 to 1.78]

5. Secondary Outcome: Locoregional Recurrences-free Survival (LRRFS)
Description: Compare locoregional recurrence-free survival (LRRFS). LRRFS is defined as the time from randomization to the date of the first event: local/regional invasive ipsilateral recurrence, contralateral invasive breast cancer, or death from any cause. Patients with second primary invasive cancers of non-breast origin or distant recurrence will be censored at the date of diagnosis. Surviving patients who are event-free will be censored at: the date of last disease assessment, or withdrawal of consent to be followed, whichever occurs first.
Time Frame: 4 years
Measure: Number; unit: percentage of patients
Arm/Group | Palbociclib Plus Endocrine Therapy (Arm A) | Endocrine Therapy Alone (Arm B)
Number analyzed (Participants) | 2884 | 2877
percentage of patients | 96.8 | 95.4
Statistical Analysis 1: Comparison: Palbociclib Plus Endocrine Therapy (Arm A) vs Endocrine Therapy Alone (Arm B); Test type: Other; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.57 to 1.23]

ADVERSE EVENTS:
Time Frame: 4 years
Description: The safety analysis is conducted in the "as-treated" population. Patients randomly assigned to the Arm A who never received Palbociclib but received endocrine therapy (N=36) were included in Arm B for the safety analyses. Thus, the safety analysis included 2841 patients who received at least one dose of Palbociclib plus endocrine therapy and 2902 patients who received endocrine therapy (which included 36 patients from Arm A who received endocrine therapy only).
Arm/Group | Palbociclib Plus Endocrine Therapy (Arm A) | Endocrine Therapy Alone (Arm B)
All-Cause Mortality (participants affected / at risk) | 99/2841 | 76/2902
Serious Adverse Events (participants affected / at risk) | 369/2841 | 229/2902
Other Adverse Events (participants affected / at risk) | 2824/2841 | 2600/2902
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Palbociclib Plus Endocrine Therapy (Arm A) (N=2841) | Endocrine Therapy Alone (Arm B) (N=2902)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 13 (13) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 4 (5) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Arteriospasm coronary (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 4 (4)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac ventricular thrombosis (Cardiac disorders) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 2 (2)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Gene mutation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Deafness unilateral (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 3 (3) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 2 (2) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Eyelid function disorder (Eye disorders) | 1 (1) | 0 (0)
Maculopathy (Eye disorders) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intussusception (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Neutropenic colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oedematous pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Peritoneal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 1 (1)
Volvulus of small bowel (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2)
Capsular contracture associated with breast implant (General disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 3 (5) | 1 (1)
Death (General disorders) | 2 (2) | 0 (0)
Disease progression (General disorders) | 1 (1) | 2 (4)
Disease recurrence (General disorders) | 1 (2) | 1 (1)
Dysplasia (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (3) | 0 (0)
Hypothermia (General disorders) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 1 (1) | 1 (1)
Implant site fibrosis (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 4 (4) | 0 (0)
Pyrexia (General disorders) | 3 (4) | 1 (1)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 3 (3) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 4 (4) | 2 (2)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Anorectal infection (Infections and infestations) | 1 (1) | 0 (0)
Appendiceal abscess (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 3 (3) | 5 (5)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Breast abscess (Infections and infestations) | 2 (2) | 1 (1)
Breast cellulitis (Infections and infestations) | 16 (17) | 10 (10)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 1 (2)
Campylobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 24 (26) | 9 (10)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 2 (2) | 4 (4)
Disseminated varicella zoster virus infection (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 3 (3)
Erysipelas (Infections and infestations) | 5 (5) | 0 (0)
Erysipelothrix sepsis (Infections and infestations) | 0 (0) | 1 (1)
Escherichia pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 4 (4) | 3 (3)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 4 (4) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Infected seroma (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 2 (2) | 3 (4)
Influenza (Infections and infestations) | 16 (16) | 2 (2)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Listeria sepsis (Infections and infestations) | 1 (2) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Mastitis (Infections and infestations) | 13 (14) | 10 (11)
Paronychia (Infections and infestations) | 1 (1) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 16 (18) | 7 (8)
Postoperative wound infection (Infections and infestations) | 1 (1) | 2 (2)
Pyelonephritis (Infections and infestations) | 2 (2) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 8 (9) | 3 (3)
Septic shock (Infections and infestations) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Skin infection (Infections and infestations) | 8 (8) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (3)
Urinary tract infection (Infections and infestations) | 8 (8) | 3 (3)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Vascular device infection (Infections and infestations) | 1 (1) | 0 (0)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 1 (2)
Viral infection (Infections and infestations) | 4 (4) | 0 (0)
Viral labyrinthitis (Infections and infestations) | 1 (1) | 0 (0)
Viral pericarditis (Infections and infestations) | 1 (1) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Wound abscess (Infections and infestations) | 2 (2) | 0 (0)
Wound infection (Infections and infestations) | 3 (4) | 4 (4)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Breast procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 3 (4)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Open fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 3 (4) | 4 (4)
Skin flap necrosis (Injury, poisoning and procedural complications) | 1 (3) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (3)
Sternal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vaginal cuff dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular access site thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 9 (9) | 5 (5)
Wrist fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Liver function test increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (5)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Acute promyelocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
B-cell small lymphocytic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 1 (1)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Intraductal papillary-mucinous carcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lymphoplasmacytoid lymphoma/immunocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Uterine leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uveal melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ageusia (Nervous system disorders) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 2 (2)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 2 (2) | 0 (0)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 1 (1)
IIIrd nerve disorder (Nervous system disorders) | 1 (1) | 0 (0)
Intercostal neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 2 (2) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 3 (3) | 0 (0)
Ruptured cerebral aneurysm (Nervous system disorders) | 1 (2) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 4 (4)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 3 (3)
VIth nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Vertigo CNS origin (Nervous system disorders) | 1 (1) | 0 (0)
Device breakage (Product Issues) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 1 (1) | 1 (3)
Device leakage (Product Issues) | 0 (0) | 1 (1)
Alcohol abuse (Psychiatric disorders) | 2 (2) | 0 (0)
Alcohol use disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
Confusional state (Psychiatric disorders) | 3 (3) | 1 (1)
Delusion (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 3 (3) | 1 (1)
Drug abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Mania (Psychiatric disorders) | 1 (1) | 0 (0)
Mental disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 2 (2) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0)
Paranoia (Psychiatric disorders) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 3 (4)
Acute kidney injury (Renal and urinary disorders) | 4 (5) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 4 (4)
Renal colic (Renal and urinary disorders) | 1 (1) | 1 (1)
Subcapsular renal haematoma (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureteric stenosis (Renal and urinary disorders) | 1 (4) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Adnexa uteri cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast calcifications (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast haematoma (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast necrosis (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Breast swelling (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cervical cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Endometrial disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Endometrial hypertrophy (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Endometrial thickening (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Vaginal haematoma (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma-chronic obstructive pulmonary disease overlap syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 5 (5)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (2)
Vocal cord dysfunction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Keloid scar (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Axillary vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Embolism (Vascular disorders) | 4 (4) | 2 (2)
Hypertensive crisis (Vascular disorders) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Palbociclib Plus Endocrine Therapy (Arm A) (N=2841) | Endocrine Therapy Alone (Arm B) (N=2902)
Agitation Mood Disturbance (Psychiatric disorders) | 0 (0) | 1 (1)
Veritgo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Agranulocytosis (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 634 (1161) | 147 (211)
Anaemia macrocytic (Blood and lymphatic system disorders) | 4 (6) | 0 (0)
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Blood disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bone marrow oedema (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 16 (16) | 0 (0)
Haematotoxicity (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Increased tendency to bruise (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 2 (6) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 397 (1798) | 64 (98)
Lymph node pain (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 6 (6) | 10 (12)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphatic disorder (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 58 (184) | 24 (40)
Macrocytosis (Blood and lymphatic system disorders) | 7 (7) | 0 (0)
Microcytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Monocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Myelosuppression (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1125 (5381) | 76 (112)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Polycythaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 195 (403) | 15 (18)
Thrombocytosis (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
White blood cell disorder (Blood and lymphatic system disorders) | 2 (4) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 4 (4) | 0 (0)
Arrhythmia (Cardiac disorders) | 2 (4) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Atrial thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 2 (2) | 5 (5)
Bundle branch block right (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 3 (3) | 3 (3)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac flutter (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac ventricular thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 2 (2)
Cardiovascular disorder (Cardiac disorders) | 1 (1) | 2 (2)
Chronic left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 3 (3)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 46 (52) | 38 (39)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Sinus arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 4 (4) | 4 (5)
Sinus tachycardia (Cardiac disorders) | 13 (14) | 12 (17)
Supraventricular tachycardia (Cardiac disorders) | 5 (5) | 1 (1)
Systolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 17 (19) | 29 (31)
Tachycardia induced cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 2 (2)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 1 (1)
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Gilbert's syndrome (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Hereditary haemochromatosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Hyper IgM syndrome (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 2 (2) | 2 (2)
Deafness (Ear and labyrinth disorders) | 4 (4) | 7 (8)
Deafness unilateral (Ear and labyrinth disorders) | 2 (3) | 2 (2)
Ear congestion (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 5 (5) | 4 (4)
Ear disorder (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 40 (43) | 11 (11)
Ear pruritus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Eustachian tube patulous (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Excessive cerumen production (Ear and labyrinth disorders) | 1 (1) | 0 (0)
External ear inflammation (Ear and labyrinth disorders) | 3 (3) | 2 (2)
External ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hyperacusis (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 9 (10) | 1 (1)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Motion sickness (Ear and labyrinth disorders) | 1 (2) | 2 (2)
Otorrhoea (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 23 (24) | 20 (20)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 74 (84) | 38 (40)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Autoimmune thyroiditis (Endocrine disorders) | 2 (2) | 4 (5)
Goitre (Endocrine disorders) | 3 (3) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 3 (3)
Hyperthyroidism (Endocrine disorders) | 5 (5) | 3 (3)
Hypothyroidism (Endocrine disorders) | 21 (22) | 41 (44)
Thyroid mass (Endocrine disorders) | 4 (4) | 7 (7)
Thyroid pain (Endocrine disorders) | 0 (0) | 1 (1)
Asthenopia (Eye disorders) | 1 (1) | 1 (1)
Blepharitis (Eye disorders) | 5 (5) | 2 (2)
Blepharospasm (Eye disorders) | 3 (3) | 1 (1)
Blindness (Eye disorders) | 1 (1) | 1 (1)
Blindness transient (Eye disorders) | 1 (1) | 1 (1)
Cataract (Eye disorders) | 16 (20) | 19 (22)
Cataract nuclear (Eye disorders) | 0 (0) | 1 (1)
Chalazion (Eye disorders) | 1 (1) | 1 (1)
Choroidal effusion (Eye disorders) | 1 (1) | 0 (0)
Conjunctival disorder (Eye disorders) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 6 (6) | 4 (4)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 0 (0)
Corneal thickening (Eye disorders) | 0 (0) | 1 (1)
Dacryostenosis acquired (Eye disorders) | 3 (3) | 0 (0)
Diplopia (Eye disorders) | 3 (3) | 2 (2)
Dry eye (Eye disorders) | 68 (75) | 42 (48)
Eye disorder (Eye disorders) | 1 (1) | 2 (2)
Eye haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Eye inflammation (Eye disorders) | 1 (1) | 1 (1)
Eye irritation (Eye disorders) | 5 (5) | 2 (2)
Eye oedema (Eye disorders) | 1 (1) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 2 (2)
Eye pruritus (Eye disorders) | 10 (11) | 5 (6)
Eye swelling (Eye disorders) | 2 (2) | 1 (1)
Eyelid cyst (Eye disorders) | 1 (1) | 0 (0)
Eyelid disorder (Eye disorders) | 1 (1) | 1 (1)
Eyelid function disorder (Eye disorders) | 1 (1) | 1 (1)
Eyelid oedema (Eye disorders) | 2 (2) | 1 (1)
Eyelid ptosis (Eye disorders) | 1 (1) | 1 (1)
Eyelids pruritus (Eye disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 3 (3) | 3 (3)
Iritis (Eye disorders) | 2 (2) | 1 (1)
Keratitis (Eye disorders) | 4 (8) | 0 (0)
Keratopathy (Eye disorders) | 1 (2) | 0 (0)
Lacrimal cyst (Eye disorders) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 96 (105) | 6 (6)
Macular degeneration (Eye disorders) | 3 (4) | 3 (3)
Macular fibrosis (Eye disorders) | 1 (1) | 0 (0)
Mydriasis (Eye disorders) | 1 (1) | 0 (0)
Neovascular age-related macular degeneration (Eye disorders) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 2 (2)
Orbital haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Orbital oedema (Eye disorders) | 1 (1) | 0 (0)
Pars plana cyst (Eye disorders) | 1 (1) | 0 (0)
Periorbital oedema (Eye disorders) | 2 (4) | 0 (0)
Periorbital swelling (Eye disorders) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 4 (4) | 3 (3)
Photopsia (Eye disorders) | 2 (2) | 2 (2)
Presbyopia (Eye disorders) | 0 (0) | 1 (1)
Punctate keratitis (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 2 (2) | 1 (1)
Retinal dystrophy (Eye disorders) | 1 (1) | 0 (0)
Retinal haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Retinal tear (Eye disorders) | 1 (1) | 2 (3)
Retinoschisis (Eye disorders) | 1 (1) | 0 (0)
Scleral cyst (Eye disorders) | 1 (1) | 0 (0)
Swelling of eyelid (Eye disorders) | 3 (3) | 0 (0)
Ulcerative keratitis (Eye disorders) | 1 (1) | 1 (1)
Uveitis (Eye disorders) | 3 (3) | 1 (2)
Vision blurred (Eye disorders) | 69 (75) | 36 (40)
Visual acuity reduced (Eye disorders) | 6 (6) | 4 (4)
Visual impairment (Eye disorders) | 19 (19) | 11 (11)
Visual snow syndrome (Eye disorders) | 1 (1) | 0 (0)
Vitreous detachment (Eye disorders) | 1 (1) | 1 (1)
Vitreous floaters (Eye disorders) | 6 (6) | 10 (10)
Xerophthalmia (Eye disorders) | 3 (3) | 1 (2)
Abdominal discomfort (Gastrointestinal disorders) | 22 (27) | 16 (16)
Abdominal distension (Gastrointestinal disorders) | 30 (36) | 33 (35)
Abdominal mass (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 153 (190) | 110 (134)
Abdominal pain lower (Gastrointestinal disorders) | 14 (14) | 16 (17)
Abdominal pain upper (Gastrointestinal disorders) | 84 (103) | 53 (61)
Abdominal rigidity (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 2 (2) | 2 (2)
Abdominal wall haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 12 (16) | 3 (3)
Anal fistula (Gastrointestinal disorders) | 3 (3) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 11 (12) | 1 (1)
Anal incontinence (Gastrointestinal disorders) | 2 (2) | 1 (1)
Anal inflammation (Gastrointestinal disorders) | 1 (2) | 0 (0)
Anal pruritus (Gastrointestinal disorders) | 1 (1) | 2 (2)
Anal skin tags (Gastrointestinal disorders) | 0 (0) | 1 (1)
Angular cheilitis (Gastrointestinal disorders) | 4 (6) | 2 (2)
Aphthous ulcer (Gastrointestinal disorders) | 16 (17) | 3 (3)
Apical granuloma (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Barrett's oesophagus (Gastrointestinal disorders) | 1 (1) | 1 (1)
Bowel movement irregularity (Gastrointestinal disorders) | 1 (1) | 0 (0)
Change of bowel habit (Gastrointestinal disorders) | 3 (3) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 4 (4) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 2 (3) | 2 (2)
Colitis (Gastrointestinal disorders) | 5 (5) | 3 (3)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 395 (485) | 172 (190)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 16 (17) | 5 (7)
Diarrhoea (Gastrointestinal disorders) | 475 (682) | 150 (194)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 5 (5) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 2 (2) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 81 (92) | 46 (49)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyschezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 137 (162) | 64 (67)
Dysphagia (Gastrointestinal disorders) | 28 (34) | 15 (16)
Enteritis (Gastrointestinal disorders) | 3 (4) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 3 (3) | 2 (3)
Epigastric discomfort (Gastrointestinal disorders) | 4 (4) | 1 (1)
Epiploic appendagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Erosive oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faeces discoloured (Gastrointestinal disorders) | 4 (4) | 0 (0)
Faeces hard (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faeces soft (Gastrointestinal disorders) | 2 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 27 (31) | 14 (15)
Food poisoning (Gastrointestinal disorders) | 3 (4) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric disorder (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 29 (32) | 9 (9)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 6 (7) | 3 (3)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 6 (7) | 3 (3)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal wall thickening (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 90 (106) | 55 (59)
Gingival bleeding (Gastrointestinal disorders) | 10 (12) | 1 (1)
Gingival discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingival oedema (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 11 (15) | 3 (3)
Gingival recession (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gingival swelling (Gastrointestinal disorders) | 2 (2) | 2 (2)
Glossitis (Gastrointestinal disorders) | 3 (4) | 2 (2)
Glossodynia (Gastrointestinal disorders) | 6 (6) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 10 (11) | 3 (3)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 7 (9) | 7 (12)
Haemorrhoids (Gastrointestinal disorders) | 43 (44) | 25 (26)
Hiatus hernia (Gastrointestinal disorders) | 4 (4) | 2 (2)
Hyperaesthesia teeth (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hypertrophic anal papilla (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 3 (4) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (2)
Intussusception (Gastrointestinal disorders) | 0 (0) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 2 (2) | 4 (4)
Large intestinal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 4 (4) | 4 (5)
Lip blister (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lip discolouration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lip disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lip dry (Gastrointestinal disorders) | 4 (4) | 1 (1)
Lip erythema (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lip pain (Gastrointestinal disorders) | 3 (3) | 0 (0)
Lip pruritus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 1 (1) | 2 (2)
Lip ulceration (Gastrointestinal disorders) | 2 (2) | 0 (0)
Loose tooth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 51 (67) | 6 (6)
Nausea (Gastrointestinal disorders) | 552 (735) | 241 (294)
Noninfective gingivitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Noninfective sialoadenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 13 (14) | 4 (5)
Oedematous pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal achalasia (Gastrointestinal disorders) | 0 (0) | 1 (2)
Oesophageal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal spasm (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 6 (8) | 3 (3)
Oral discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral dysaesthesia (Gastrointestinal disorders) | 5 (5) | 0 (0)
Oral mucosal blistering (Gastrointestinal disorders) | 1 (3) | 0 (0)
Oral pain (Gastrointestinal disorders) | 49 (61) | 6 (6)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Paraesthesia oral (Gastrointestinal disorders) | 4 (5) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 3 (3) | 2 (2)
Proctalgia (Gastrointestinal disorders) | 6 (6) | 1 (1)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ranula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 20 (21) | 12 (13)
Rectal lesion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal tenesmus (Gastrointestinal disorders) | 1 (2) | 2 (2)
Rectal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Reflux gastritis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Salivary duct inflammation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Salivary gland calculus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 280 (428) | 21 (23)
Swollen tongue (Gastrointestinal disorders) | 1 (1) | 2 (2)
Teeth brittle (Gastrointestinal disorders) | 1 (1) | 1 (1)
Tongue coated (Gastrointestinal disorders) | 2 (2) | 0 (0)
Tongue geographic (Gastrointestinal disorders) | 1 (2) | 0 (0)
Tongue ulceration (Gastrointestinal disorders) | 7 (7) | 0 (0)
Tooth disorder (Gastrointestinal disorders) | 2 (2) | 0 (0)
Tooth loss (Gastrointestinal disorders) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 35 (39) | 17 (18)
Umbilical hernia (Gastrointestinal disorders) | 2 (2) | 2 (2)
Volvulus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 219 (278) | 91 (120)
Acute phase reaction (General disorders) | 0 (0) | 1 (1)
Adverse drug reaction (General disorders) | 1 (1) | 2 (2)
Application site coldness (General disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 274 (468) | 153 (193)
Axillary pain (General disorders) | 43 (44) | 48 (55)
Capsular contracture associated with breast implant (General disorders) | 2 (2) | 2 (2)
Capsular contracture associated with implant (General disorders) | 0 (0) | 1 (1)
Catheter site inflammation (General disorders) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 6 (7)
Catheter site pruritus (General disorders) | 0 (0) | 1 (1)
Catheter site scab (General disorders) | 1 (1) | 0 (0)
Catheter site thrombosis (General disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 37 (42) | 22 (24)
Chest pain (General disorders) | 56 (64) | 51 (54)
Chills (General disorders) | 70 (78) | 17 (17)
Complication associated with device (General disorders) | 1 (1) | 0 (0)
Cyst (General disorders) | 7 (7) | 7 (7)
Decreased activity (General disorders) | 1 (1) | 0 (0)
Discomfort (General disorders) | 7 (7) | 7 (7)
Early satiety (General disorders) | 1 (1) | 0 (0)
Exercise tolerance decreased (General disorders) | 1 (1) | 2 (2)
Face oedema (General disorders) | 5 (5) | 4 (4)
Facial pain (General disorders) | 4 (4) | 4 (4)
Fat necrosis (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 1163 (1869) | 560 (714)
Feeling abnormal (General disorders) | 3 (3) | 3 (3)
Feeling cold (General disorders) | 3 (3) | 2 (2)
Feeling hot (General disorders) | 1 (1) | 0 (0)
Feeling jittery (General disorders) | 1 (1) | 0 (0)
Fibrosis (General disorders) | 1 (1) | 3 (3)
Gait disturbance (General disorders) | 6 (6) | 6 (6)
General physical health deterioration (General disorders) | 6 (7) | 2 (2)
Granuloma (General disorders) | 2 (2) | 1 (1)
Hernia pain (General disorders) | 0 (0) | 2 (2)
Hyperthermia (General disorders) | 1 (1) | 0 (0)
Hypertrophy (General disorders) | 1 (1) | 1 (1)
Hypothermia (General disorders) | 2 (2) | 0 (0)
Illness (General disorders) | 4 (5) | 2 (2)
Impaired healing (General disorders) | 14 (14) | 5 (6)
Implant site pain (General disorders) | 1 (2) | 3 (3)
Induration (General disorders) | 0 (0) | 1 (1)
Inflammation (General disorders) | 3 (3) | 2 (2)
Influenza like illness (General disorders) | 166 (205) | 90 (108)
Injection site pain (General disorders) | 0 (0) | 1 (1)
Injection site phlebitis (General disorders) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 1 (1) | 1 (1)
Localised oedema (General disorders) | 16 (16) | 10 (11)
Malaise (General disorders) | 32 (34) | 11 (16)
Mass (General disorders) | 5 (5) | 3 (3)
Mucosal disorder (General disorders) | 1 (1) | 0 (0)
Mucosal dryness (General disorders) | 11 (12) | 14 (15)
Mucosal haemorrhage (General disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 206 (362) | 10 (10)
Mucosal pain (General disorders) | 1 (1) | 0 (0)
Mucosal toxicity (General disorders) | 1 (1) | 0 (0)
Necrosis (General disorders) | 1 (1) | 1 (1)
Nodule (General disorders) | 4 (6) | 5 (6)
Non-cardiac chest pain (General disorders) | 24 (29) | 29 (33)
Oedema (General disorders) | 27 (35) | 25 (29)
Oedema peripheral (General disorders) | 178 (218) | 121 (137)
Pain (General disorders) | 107 (122) | 94 (102)
Pelvic mass (General disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 55 (61) | 33 (36)
Polyp (General disorders) | 2 (2) | 1 (2)
Pyrexia (General disorders) | 205 (251) | 83 (92)
Sensitivity to weather change (General disorders) | 1 (1) | 1 (1)
Suprapubic pain (General disorders) | 0 (0) | 1 (1)
Swelling (General disorders) | 13 (17) | 9 (10)
Swelling face (General disorders) | 3 (3) | 2 (2)
Temperature intolerance (General disorders) | 6 (6) | 1 (1)
Temperature regulation disorder (General disorders) | 2 (2) | 0 (0)
Tenderness (General disorders) | 10 (10) | 3 (3)
Thirst (General disorders) | 1 (1) | 3 (3)
Unevaluable event (General disorders) | 9 (9) | 4 (4)
Vessel puncture site pain (General disorders) | 1 (1) | 0 (0)
Xerosis (General disorders) | 6 (7) | 2 (2)
Biliary colic (Hepatobiliary disorders) | 2 (2) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 8 (8) | 4 (4)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 7 (7) | 8 (9)
Gallbladder polyp (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic cyst (Hepatobiliary disorders) | 1 (1) | 2 (2)
Hepatic lesion (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic pain (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 9 (9) | 9 (9)
Hepatitis toxic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatocellular injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 (3) | 5 (12)
Hypertransaminasaemia (Hepatobiliary disorders) | 2 (3) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver tenderness (Hepatobiliary disorders) | 1 (1) | 0 (0)
Porcelain gallbladder (Hepatobiliary disorders) | 1 (1) | 1 (1)
Steatohepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Allergy to arthropod bite (Immune system disorders) | 1 (1) | 1 (1)
Allergy to vaccine (Immune system disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 5 (6) | 2 (2)
Food allergy (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 16 (18) | 4 (4)
Immune system disorder (Immune system disorders) | 0 (0) | 2 (3)
Mite allergy (Immune system disorders) | 0 (0) | 1 (1)
Multiple allergies (Immune system disorders) | 2 (2) | 3 (3)
Perfume sensitivity (Immune system disorders) | 0 (0) | 1 (1)
Sarcoidosis (Immune system disorders) | 2 (2) | 0 (0)
Seasonal allergy (Immune system disorders) | 19 (20) | 10 (11)
Abdominal infection (Infections and infestations) | 1 (1) | 1 (1)
Abscess (Infections and infestations) | 3 (4) | 2 (2)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Abscess neck (Infections and infestations) | 1 (1) | 0 (0)
Abscess oral (Infections and infestations) | 4 (4) | 1 (1)
Acarodermatitis (Infections and infestations) | 2 (2) | 0 (0)
Acute sinusitis (Infections and infestations) | 2 (2) | 3 (4)
Anal abscess (Infections and infestations) | 2 (2) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 2 (2)
Arthritis infective (Infections and infestations) | 1 (1) | 0 (0)
Babesiosis (Infections and infestations) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Bacterial vaginosis (Infections and infestations) | 2 (2) | 4 (4)
Bacterial vulvovaginitis (Infections and infestations) | 0 (0) | 1 (1)
Bacteriuria (Infections and infestations) | 0 (0) | 1 (1)
Bartholin's abscess (Infections and infestations) | 0 (0) | 1 (1)
Beta haemolytic streptococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Blastocystis infection (Infections and infestations) | 0 (0) | 1 (1)
Blister infected (Infections and infestations) | 1 (1) | 0 (0)
Breast abscess (Infections and infestations) | 2 (2) | 0 (0)
Breast cellulitis (Infections and infestations) | 17 (22) | 15 (15)
Bronchitis (Infections and infestations) | 68 (85) | 56 (60)
Bronchitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis viral (Infections and infestations) | 2 (2) | 0 (0)
COVID-19 (Infections and infestations) | 3 (3) | 2 (2)
Candida infection (Infections and infestations) | 15 (18) | 6 (6)
Catheter site pustule (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 53 (66) | 31 (38)
Cervicitis (Infections and infestations) | 1 (1) | 0 (0)
Cervicitis human papilloma virus (Infections and infestations) | 1 (1) | 0 (0)
Chest wall abscess (Infections and infestations) | 0 (0) | 1 (1)
Chronic hepatitis C (Infections and infestations) | 1 (1) | 0 (0)
Chronic sinusitis (Infections and infestations) | 2 (2) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 36 (37) | 27 (28)
Conjunctivitis bacterial (Infections and infestations) | 1 (1) | 1 (1)
Conjunctivitis viral (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 30 (34) | 29 (33)
Dacryocystitis (Infections and infestations) | 1 (1) | 0 (0)
Demodicidosis (Infections and infestations) | 1 (1) | 0 (0)
Dengue fever (Infections and infestations) | 0 (0) | 1 (1)
Dermatophytosis (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 3 (4)
Diverticulitis (Infections and infestations) | 7 (8) | 2 (2)
Ear infection (Infections and infestations) | 20 (23) | 10 (11)
Ear infection fungal (Infections and infestations) | 0 (0) | 1 (1)
Endometritis (Infections and infestations) | 1 (2) | 0 (0)
Enteritis infectious (Infections and infestations) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 2 (2) | 1 (1)
Epstein-Barr virus infection (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 9 (11) | 3 (3)
Erythema migrans (Infections and infestations) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 17 (20) | 7 (8)
Eyelid infection (Infections and infestations) | 1 (1) | 0 (0)
Febrile infection (Infections and infestations) | 1 (1) | 1 (1)
Folliculitis (Infections and infestations) | 10 (12) | 9 (9)
Fungal infection (Infections and infestations) | 16 (18) | 9 (9)
Fungal skin infection (Infections and infestations) | 6 (6) | 6 (7)
Furuncle (Infections and infestations) | 3 (5) | 0 (0)
Gastroenteritis (Infections and infestations) | 46 (51) | 20 (21)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis salmonella (Infections and infestations) | 1 (2) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 18 (19) | 10 (10)
Gastrointestinal bacterial overgrowth (Infections and infestations) | 1 (1) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 5 (5) | 4 (4)
Gastrointestinal viral infection (Infections and infestations) | 4 (4) | 0 (0)
Genital herpes (Infections and infestations) | 3 (4) | 3 (3)
Genital herpes simplex (Infections and infestations) | 1 (1) | 0 (0)
Gingival abscess (Infections and infestations) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 6 (7) | 9 (9)
Haemophilus infection (Infections and infestations) | 0 (0) | 1 (1)
Haemorrhoid infection (Infections and infestations) | 1 (1) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 1 (1)
Helicobacter gastritis (Infections and infestations) | 1 (1) | 1 (1)
Helicobacter infection (Infections and infestations) | 6 (6) | 4 (4)
Herpes ophthalmic (Infections and infestations) | 0 (0) | 2 (2)
Herpes simplex (Infections and infestations) | 12 (13) | 4 (4)
Herpes simplex reactivation (Infections and infestations) | 1 (1) | 0 (0)
Herpes virus infection (Infections and infestations) | 9 (10) | 3 (6)
Herpes zoster (Infections and infestations) | 52 (57) | 50 (53)
Hordeolum (Infections and infestations) | 6 (6) | 8 (8)
Incision site cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Infected bite (Infections and infestations) | 4 (4) | 1 (1)
Infected cyst (Infections and infestations) | 0 (0) | 1 (1)
Infected dermal cyst (Infections and infestations) | 1 (1) | 2 (2)
Infected seroma (Infections and infestations) | 1 (1) | 2 (4)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 17 (18) | 10 (11)
Infection parasitic (Infections and infestations) | 1 (1) | 0 (0)
Infective tenosynovitis (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 102 (109) | 45 (48)
Kidney infection (Infections and infestations) | 1 (1) | 1 (1)
Labyrinthitis (Infections and infestations) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 21 (22) | 5 (5)
Laryngitis viral (Infections and infestations) | 1 (1) | 0 (0)
Lip infection (Infections and infestations) | 8 (8) | 3 (3)
Localised infection (Infections and infestations) | 7 (8) | 4 (4)
Lower respiratory tract infection (Infections and infestations) | 36 (49) | 20 (21)
Lower respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Lyme disease (Infections and infestations) | 4 (4) | 2 (2)
Lymph gland infection (Infections and infestations) | 0 (0) | 2 (2)
Lymphangitis (Infections and infestations) | 4 (4) | 2 (3)
Mastitis (Infections and infestations) | 29 (43) | 43 (47)
Mucosal infection (Infections and infestations) | 6 (8) | 3 (3)
Nail infection (Infections and infestations) | 5 (5) | 5 (7)
Nasal abscess (Infections and infestations) | 3 (4) | 0 (0)
Nasal herpes (Infections and infestations) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 210 (275) | 127 (157)
Nipple infection (Infections and infestations) | 1 (1) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Oesophageal infection (Infections and infestations) | 1 (1) | 0 (0)
Onychomycosis (Infections and infestations) | 8 (9) | 7 (7)
Oral candidiasis (Infections and infestations) | 12 (13) | 4 (4)
Oral fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 65 (88) | 16 (17)
Oral infection (Infections and infestations) | 4 (4) | 2 (2)
Otitis externa (Infections and infestations) | 6 (6) | 3 (3)
Otitis media (Infections and infestations) | 19 (22) | 5 (5)
Papilloma viral infection (Infections and infestations) | 1 (1) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 1 (1)
Parasitic gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Paronychia (Infections and infestations) | 9 (9) | 8 (8)
Parotitis (Infections and infestations) | 1 (1) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 1 (1) | 0 (0)
Pericoronitis (Infections and infestations) | 1 (1) | 0 (0)
Perineal abscess (Infections and infestations) | 1 (1) | 1 (1)
Periodontitis (Infections and infestations) | 3 (4) | 1 (1)
Periorbital cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Periorbital infection (Infections and infestations) | 1 (1) | 0 (0)
Peripheral nerve infection (Infections and infestations) | 1 (1) | 0 (0)
Periumbilical abscess (Infections and infestations) | 1 (1) | 0 (0)
Pertussis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 50 (63) | 19 (20)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 1 (1)
Pilonidal cyst (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 38 (42) | 35 (37)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 1 (1)
Post procedural cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 8 (8) | 3 (3)
Psoas abscess (Infections and infestations) | 1 (1) | 0 (0)
Pulpitis dental (Infections and infestations) | 2 (3) | 2 (2)
Pustule (Infections and infestations) | 3 (3) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 3 (3)
Rash pustular (Infections and infestations) | 12 (13) | 4 (5)
Respiratory tract infection (Infections and infestations) | 52 (73) | 31 (35)
Respiratory tract infection viral (Infections and infestations) | 3 (4) | 3 (3)
Rhinitis (Infections and infestations) | 36 (46) | 12 (13)
Sialoadenitis (Infections and infestations) | 1 (1) | 0 (0)
Sinobronchitis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 105 (132) | 61 (74)
Skin candida (Infections and infestations) | 2 (2) | 3 (3)
Skin infection (Infections and infestations) | 63 (85) | 29 (31)
Soft tissue infection (Infections and infestations) | 2 (2) | 3 (3)
Sputum purulent (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 2 (3)
Streptococcal infection (Infections and infestations) | 1 (3) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Suspected COVID-19 (Infections and infestations) | 1 (1) | 1 (1)
Tinea infection (Infections and infestations) | 0 (0) | 1 (1)
Tinea pedis (Infections and infestations) | 4 (4) | 1 (1)
Tinea versicolour (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 9 (10) | 10 (10)
Tooth abscess (Infections and infestations) | 14 (16) | 7 (8)
Tooth infection (Infections and infestations) | 26 (30) | 21 (21)
Toxoplasmosis (Infections and infestations) | 0 (0) | 1 (1)
Tracheitis (Infections and infestations) | 7 (8) | 0 (0)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 304 (390) | 185 (229)
Urethritis (Infections and infestations) | 1 (2) | 1 (2)
Urinary tract infection (Infections and infestations) | 234 (320) | 145 (204)
Urinary tract infection viral (Infections and infestations) | 1 (1) | 1 (1)
Vaginal infection (Infections and infestations) | 27 (28) | 18 (21)
Varicella (Infections and infestations) | 0 (0) | 1 (1)
Vascular device infection (Infections and infestations) | 1 (1) | 1 (1)
Vestibulitis (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 28 (30) | 18 (18)
Viral skin infection (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 7 (7) | 5 (6)
Vulval cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Vulvitis (Infections and infestations) | 2 (2) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 15 (17) | 3 (3)
Vulvovaginal human papilloma virus infection (Infections and infestations) | 1 (1) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 8 (8) | 12 (13)
Wound infection (Infections and infestations) | 14 (16) | 7 (8)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Ankle fracture (Injury, poisoning and procedural complications) | 10 (11) | 13 (13)
Arthropod bite (Injury, poisoning and procedural complications) | 22 (24) | 11 (11)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Axillary web syndrome (Injury, poisoning and procedural complications) | 14 (15) | 5 (5)
Back injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Breast injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Breast procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chillblains (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 4 (6)
Compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 95 (108) | 37 (43)
Corneal abrasion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Epicondylitis (Injury, poisoning and procedural complications) | 5 (6) | 3 (3)
Exposure to toxic agent (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 57 (68) | 40 (49)
Fibula fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 10 (10) | 16 (17)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Fractured coccyx (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fractured sacrum (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastroparesis postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hair injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (2) | 4 (4)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Heat stroke (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 3 (3) | 5 (5)
Iliotibial band syndrome (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Incision site complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Incision site erythema (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Incision site fibrosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Incision site pain (Injury, poisoning and procedural complications) | 18 (21) | 17 (19)
Incision site pruritus (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 2 (3) | 2 (2)
Joint injury (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 2 (2) | 5 (6)
Ligament sprain (Injury, poisoning and procedural complications) | 12 (12) | 10 (10)
Limb injury (Injury, poisoning and procedural complications) | 8 (8) | 4 (4)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Median nerve injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 5 (6) | 7 (7)
Mouth injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Mucosal excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle rupture (Injury, poisoning and procedural complications) | 1 (2) | 3 (3)
Muscle strain (Injury, poisoning and procedural complications) | 6 (6) | 4 (4)
Musculoskeletal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Musculoskeletal procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Nail injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Nerve injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Post procedural constipation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural discomfort (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Post procedural inflammation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post procedural oedema (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural swelling (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (4)
Postpericardiotomy syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 48 (58) | 45 (55)
Procedural site reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural vomiting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pulmonary radiation injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Radiation associated pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radiation fibrosis (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Radiation fibrosis - lung (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Radiation neuropathy (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 6 (6) | 6 (7)
Radiation skin injury (Injury, poisoning and procedural complications) | 12 (15) | 20 (20)
Radius fracture (Injury, poisoning and procedural complications) | 7 (7) | 6 (6)
Rectal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 10 (10) | 12 (13)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Scar (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 24 (28) | 36 (46)
Skin abrasion (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Skin flap necrosis (Injury, poisoning and procedural complications) | 1 (3) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 4 (4) | 4 (4)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 5 (8)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stress fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Suture related complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Synovial rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 5 (5)
Thermal burn (Injury, poisoning and procedural complications) | 6 (6) | 8 (10)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Tooth fracture (Injury, poisoning and procedural complications) | 9 (9) | 3 (4)
Traumatic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 7 (7) | 5 (7)
Vascular access site thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 12 (12) | 4 (5)
Wound complication (Injury, poisoning and procedural complications) | 19 (21) | 3 (3)
Wound decomposition (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 16 (19) | 7 (7)
Wound secretion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 9 (9) | 10 (10)
AST/ALT ratio abnormal (Investigations) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0)
Alanine aminotransferase (Investigations) | 0 (0) | 1 (1)
Alanine aminotransferase decreased (Investigations) | 5 (6) | 4 (4)
Alanine aminotransferase increased (Investigations) | 212 (345) | 138 (175)
Albumin globulin ratio decreased (Investigations) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 2 (2)
Anion gap decreased (Investigations) | 1 (1) | 0 (0)
Anion gap increased (Investigations) | 5 (6) | 1 (1)
Antimitochondrial antibody positive (Investigations) | 1 (1) | 0 (0)
Antinuclear antibody increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase (Investigations) | 2 (2) | 1 (1)
Aspartate aminotransferase decreased (Investigations) | 6 (6) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 210 (288) | 114 (151)
Bacterial test (Investigations) | 0 (0) | 2 (2)
Basophil count increased (Investigations) | 5 (7) | 0 (0)
Bilirubin conjugated decreased (Investigations) | 0 (0) | 3 (5)
Biopsy skin (Investigations) | 0 (0) | 1 (1)
Blood 1,25-dihydroxycholecalciferol decreased (Investigations) | 0 (0) | 1 (1)
Blood albumin decreased (Investigations) | 5 (6) | 8 (9)
Blood albumin increased (Investigations) | 2 (2) | 1 (1)
Blood alkaline phosphatase (Investigations) | 5 (7) | 2 (2)
Blood alkaline phosphatase decreased (Investigations) | 6 (8) | 4 (4)
Blood alkaline phosphatase increased (Investigations) | 75 (91) | 98 (127)
Blood bicarbonate increased (Investigations) | 0 (0) | 1 (1)
Blood bilirubin (Investigations) | 1 (1) | 1 (1)
Blood bilirubin abnormal (Investigations) | 0 (0) | 2 (2)
Blood bilirubin decreased (Investigations) | 0 (0) | 2 (2)
Blood bilirubin increased (Investigations) | 29 (47) | 28 (41)
Blood calcium decreased (Investigations) | 6 (8) | 2 (3)
Blood calcium increased (Investigations) | 1 (1) | 3 (4)
Blood chloride decreased (Investigations) | 0 (0) | 3 (5)
Blood chloride increased (Investigations) | 4 (4) | 2 (2)
Blood cholesterol increased (Investigations) | 21 (22) | 47 (51)
Blood creatine increased (Investigations) | 1 (1) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 4 (4) | 0 (0)
Blood creatinine decreased (Investigations) | 5 (5) | 3 (4)
Blood creatinine increased (Investigations) | 91 (133) | 50 (80)
Blood culture positive (Investigations) | 1 (1) | 0 (0)
Blood folate decreased (Investigations) | 2 (2) | 0 (0)
Blood glucose decreased (Investigations) | 2 (4) | 2 (2)
Blood glucose increased (Investigations) | 17 (24) | 25 (30)
Blood iron decreased (Investigations) | 1 (1) | 1 (1)
Blood ketone body (Investigations) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 8 (8) | 0 (0)
Blood magnesium decreased (Investigations) | 3 (3) | 4 (4)
Blood phosphorus decreased (Investigations) | 0 (0) | 2 (2)
Blood phosphorus increased (Investigations) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 8 (9) | 1 (1)
Blood potassium increased (Investigations) | 2 (4) | 2 (2)
Blood pressure diastolic increased (Investigations) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 3 (3) | 5 (8)
Blood pressure systolic increased (Investigations) | 1 (1) | 1 (1)
Blood sodium decreased (Investigations) | 1 (1) | 3 (4)
Blood sodium increased (Investigations) | 0 (0) | 3 (3)
Blood testosterone decreased (Investigations) | 0 (0) | 1 (1)
Blood thyroid stimulating hormone decreased (Investigations) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 2 (2) | 2 (2)
Blood triglycerides increased (Investigations) | 6 (6) | 7 (10)
Blood urea decreased (Investigations) | 2 (3) | 2 (3)
Blood urea increased (Investigations) | 11 (15) | 8 (11)
Blood urea nitrogen/creatinine ratio (Investigations) | 2 (4) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 6 (6)
Blood urine present (Investigations) | 2 (2) | 0 (0)
Body temperature increased (Investigations) | 2 (2) | 2 (2)
Bone density decreased (Investigations) | 1 (1) | 0 (0)
Brain natriuretic peptide increased (Investigations) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 4 (4) | 0 (0)
Carbon dioxide abnormal (Investigations) | 3 (3) | 1 (1)
Carbon dioxide decreased (Investigations) | 3 (3) | 2 (2)
Carbon dioxide increased (Investigations) | 2 (2) | 3 (3)
Cardiac murmur (Investigations) | 4 (4) | 2 (2)
Carotid bruit (Investigations) | 1 (1) | 0 (0)
Coagulation time prolonged (Investigations) | 1 (1) | 0 (0)
Colonoscopy abnormal (Investigations) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 4 (5) | 3 (3)
Electrocardiogram QT prolonged (Investigations) | 2 (2) | 0 (0)
Eosinophil count increased (Investigations) | 2 (2) | 2 (3)
Eosinophil percentage decreased (Investigations) | 0 (0) | 1 (1)
Eosinophil percentage increased (Investigations) | 0 (0) | 2 (2)
Fibrin D dimer increased (Investigations) | 0 (0) | 1 (1)
Gamma-glutamyltransferase (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 18 (35) | 21 (35)
Glomerular filtration rate decreased (Investigations) | 6 (11) | 1 (1)
Glomerular filtration rate increased (Investigations) | 1 (2) | 0 (0)
Glycosylated haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Glycosylated haemoglobin increased (Investigations) | 15 (18) | 20 (22)
Granulocyte count decreased (Investigations) | 1 (2) | 0 (0)
Granulocyte count increased (Investigations) | 1 (1) | 0 (0)
Haematocrit decreased (Investigations) | 28 (41) | 6 (7)
Haemoglobin decreased (Investigations) | 42 (79) | 12 (15)
Haemoglobin increased (Investigations) | 0 (0) | 2 (2)
Heart rate decreased (Investigations) | 1 (1) | 0 (0)
Heart rate increased (Investigations) | 4 (6) | 2 (3)
Heart rate irregular (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 7 (9) | 5 (5)
High density lipoprotein decreased (Investigations) | 3 (3) | 0 (0)
Influenza A virus test positive (Investigations) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 1 (2) | 2 (5)
Intestinal transit time abnormal (Investigations) | 1 (1) | 0 (0)
Intraocular pressure increased (Investigations) | 1 (1) | 2 (2)
Liver function test abnormal (Investigations) | 1 (1) | 1 (1)
Liver function test increased (Investigations) | 4 (4) | 8 (8)
Low density lipoprotein increased (Investigations) | 1 (1) | 0 (0)
Lymph node palpable (Investigations) | 0 (0) | 1 (1)
Lymphocyte count (Investigations) | 1 (2) | 1 (1)
Lymphocyte count decreased (Investigations) | 317 (926) | 100 (161)
Lymphocyte count increased (Investigations) | 7 (7) | 1 (2)
Lymphocyte percentage increased (Investigations) | 1 (2) | 0 (0)
Mean cell haemoglobin concentration (Investigations) | 0 (0) | 1 (1)
Mean cell haemoglobin concentration abnormal (Investigations) | 0 (0) | 1 (1)
Mean cell haemoglobin concentration decreased (Investigations) | 1 (1) | 0 (0)
Mean cell haemoglobin concentration increased (Investigations) | 3 (3) | 0 (0)
Mean cell haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Mean cell haemoglobin increased (Investigations) | 11 (14) | 1 (1)
Mean cell volume (Investigations) | 1 (1) | 0 (0)
Mean cell volume abnormal (Investigations) | 8 (8) | 0 (0)
Mean cell volume decreased (Investigations) | 2 (2) | 0 (0)
Mean cell volume increased (Investigations) | 14 (17) | 1 (1)
Mean platelet volume decreased (Investigations) | 5 (6) | 2 (3)
Mean platelet volume increased (Investigations) | 1 (2) | 0 (0)
Monocyte count decreased (Investigations) | 13 (24) | 1 (1)
Monocyte count increased (Investigations) | 8 (9) | 1 (1)
Monocyte percentage decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil count (Investigations) | 9 (13) | 0 (0)
Neutrophil count abnormal (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1344 (6144) | 67 (109)
Neutrophil count increased (Investigations) | 4 (5) | 6 (6)
Neutrophil percentage decreased (Investigations) | 0 (0) | 1 (2)
Non-high-density lipoprotein cholesterol increased (Investigations) | 1 (1) | 1 (1)
Occult blood positive (Investigations) | 0 (0) | 1 (1)
Pancreatic enzymes decreased (Investigations) | 1 (1) | 0 (0)
Physical examination abnormal (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 436 (850) | 35 (50)
Platelet count increased (Investigations) | 7 (7) | 2 (2)
Prostatic specific antigen increased (Investigations) | 1 (1) | 0 (0)
Protein total abnormal (Investigations) | 1 (1) | 0 (0)
Protein total decreased (Investigations) | 5 (5) | 8 (10)
Protein total increased (Investigations) | 0 (0) | 1 (1)
Red blood cell count decreased (Investigations) | 35 (49) | 7 (7)
Red blood cell count increased (Investigations) | 1 (1) | 0 (0)
Red blood cell sedimentation rate increased (Investigations) | 1 (1) | 1 (1)
Red cell distribution width decreased (Investigations) | 1 (1) | 0 (0)
Red cell distribution width increased (Investigations) | 13 (14) | 1 (1)
Rheumatoid factor increased (Investigations) | 1 (1) | 0 (0)
Smear cervix abnormal (Investigations) | 0 (0) | 1 (1)
Specific gravity urine increased (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 7 (8) | 7 (7)
Troponin I increased (Investigations) | 1 (1) | 1 (1)
Urine analysis abnormal (Investigations) | 1 (1) | 0 (0)
Urine leukocyte esterase (Investigations) | 0 (0) | 1 (1)
Vitamin B12 decreased (Investigations) | 4 (4) | 1 (1)
Vitamin D decreased (Investigations) | 9 (9) | 13 (13)
Weight decreased (Investigations) | 44 (48) | 29 (40)
Weight increased (Investigations) | 116 (155) | 136 (162)
White blood cell count (Investigations) | 3 (3) | 0 (0)
White blood cell count decreased (Investigations) | 1187 (5122) | 155 (242)
White blood cell count increased (Investigations) | 1 (1) | 4 (4)
White blood cells urine (Investigations) | 1 (1) | 0 (0)
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Appetite disorder (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 151 (176) | 73 (87)
Dehydration (Metabolism and nutrition disorders) | 17 (18) | 5 (5)
Diabetes mellitus (Metabolism and nutrition disorders) | 3 (3) | 6 (6)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dyslipidaemia (Metabolism and nutrition disorders) | 2 (2) | 8 (9)
Fluid retention (Metabolism and nutrition disorders) | 5 (5) | 10 (11)
Folate deficiency (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Food craving (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 3 (3) | 6 (7)
Gout (Metabolism and nutrition disorders) | 5 (6) | 4 (4)
Hyperalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 45 (59) | 44 (61)
Hyperchloraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 8 (8) | 23 (30)
Hyperglycaemia (Metabolism and nutrition disorders) | 119 (185) | 95 (141)
Hyperkalaemia (Metabolism and nutrition disorders) | 29 (36) | 35 (35)
Hyperlipidaemia (Metabolism and nutrition disorders) | 6 (6) | 9 (9)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 29 (32) | 35 (39)
Hyperphagia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 13 (15) | 14 (17)
Hyperuricaemia (Metabolism and nutrition disorders) | 5 (6) | 10 (14)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 43 (63) | 28 (40)
Hypocalcaemia (Metabolism and nutrition disorders) | 47 (69) | 30 (35)
Hypochloraemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 24 (24) | 17 (18)
Hypokalaemia (Metabolism and nutrition disorders) | 93 (140) | 53 (69)
Hypomagnesaemia (Metabolism and nutrition disorders) | 22 (23) | 8 (10)
Hyponatraemia (Metabolism and nutrition disorders) | 50 (57) | 36 (46)
Hypophosphataemia (Metabolism and nutrition disorders) | 15 (20) | 7 (9)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypovitaminosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 3 (3) | 6 (6)
Iron deficiency (Metabolism and nutrition disorders) | 1 (2) | 3 (3)
Lipoedema (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 3 (7) | 0 (0)
Polydipsia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Tetany (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (4) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Vitamin B complex deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 6 (6) | 2 (2)
Vitamin D deficiency (Metabolism and nutrition disorders) | 29 (29) | 25 (26)
Weight loss poor (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1087 (1650) | 1305 (2034)
Arthritis (Musculoskeletal and connective tissue disorders) | 25 (28) | 33 (41)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (2)
Axillary mass (Musculoskeletal and connective tissue disorders) | 6 (6) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 311 (369) | 287 (346)
Bone disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone loss (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 80 (93) | 87 (97)
Bursitis (Musculoskeletal and connective tissue disorders) | 13 (13) | 14 (16)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest wall haematoma (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest wall mass (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Chest wall necrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chondromalacia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 7 (8) | 9 (9)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2)
Enthesopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 1 (1)
Fistula (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 23 (25) | 12 (14)
Foot deformity (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Groin pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 8 (8)
Hand deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Interspinous osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 7 (7) | 8 (8)
Jaw cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint ankylosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4)
Joint contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Joint effusion (Musculoskeletal and connective tissue disorders) | 7 (8) | 1 (1)
Joint instability (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint noise (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 33 (36) | 29 (34)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 58 (63) | 49 (52)
Joint swelling (Musculoskeletal and connective tissue disorders) | 20 (23) | 15 (20)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 8 (10) | 12 (13)
Limb mass (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Lupus-like syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Mandibular mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Medial tibial stress syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 6 (7) | 5 (6)
Muscle discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 193 (229) | 124 (131)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 3 (4) | 12 (12)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (4)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 45 (51) | 29 (32)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 99 (117) | 85 (92)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 16 (23) | 20 (25)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (6)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 65 (93) | 81 (107)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 40 (47) | 64 (71)
Myalgia (Musculoskeletal and connective tissue disorders) | 250 (315) | 235 (276)
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 69 (73) | 72 (78)
Nodal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 18 (19) | 27 (30)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Osteopenia (Musculoskeletal and connective tissue disorders) | 60 (60) | 70 (70)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 75 (75) | 90 (91)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 265 (347) | 280 (349)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 21 (22) | 12 (14)
Periarthritis (Musculoskeletal and connective tissue disorders) | 7 (7) | 10 (11)
Periostitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Plantar fascial fibromatosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 16 (17) | 16 (17)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pubic pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 3 (3) | 12 (12)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Soft tissue swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (6)
Spinal pain (Musculoskeletal and connective tissue disorders) | 8 (10) | 10 (11)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Spinal synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 3 (3) | 10 (11)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Systemic scleroderma (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Tendon calcification (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendon discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5)
Tendon pain (Musculoskeletal and connective tissue disorders) | 5 (7) | 2 (2)
Tendon sheath disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 28 (32) | 28 (35)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (6)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 9 (13) | 9 (10)
Torticollis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 28 (35) | 28 (29)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Wrist deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 14 (15)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 4 (4)
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Borderline serous tumour of ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Hair follicle tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hypergammaglobulinaemia benign monoclonal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Intraductal papillary-mucinous carcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Keratinising squamous cell carcinoma of nasopharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 6 (8)
Lipoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (9) | 6 (6)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mucinous adenocarcinoma of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oral fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal hamartoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Sarcomatoid mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Serous cystadenocarcinoma ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (6) | 3 (3)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tendon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 8 (8)
Vulval neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Vulvovaginal warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ageusia (Nervous system disorders) | 5 (5) | 0 (0)
Akathisia (Nervous system disorders) | 1 (1) | 1 (1)
Allodynia (Nervous system disorders) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 24 (24) | 21 (23)
Anosmia (Nervous system disorders) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 2 (2) | 3 (4)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Auditory nerve disorder (Nervous system disorders) | 1 (1) | 0 (0)
Aura (Nervous system disorders) | 1 (1) | 0 (0)
Autonomic nervous system imbalance (Nervous system disorders) | 1 (1) | 0 (0)
Balance disorder (Nervous system disorders) | 5 (5) | 4 (4)
Brachial plexopathy (Nervous system disorders) | 0 (0) | 2 (2)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0)
Burning sensation (Nervous system disorders) | 4 (4) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 21 (25) | 31 (35)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 1 (1)
Cerebrovascular disorder (Nervous system disorders) | 1 (1) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 2 (2) | 0 (0)
Cognitive disorder (Nervous system disorders) | 34 (41) | 20 (22)
Complex regional pain syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 1 (1) | 0 (0)
Demyelination (Nervous system disorders) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 1 (1)
Disturbance in attention (Nervous system disorders) | 33 (38) | 22 (22)
Dizziness (Nervous system disorders) | 248 (306) | 169 (190)
Dizziness postural (Nervous system disorders) | 4 (4) | 2 (2)
Drooling (Nervous system disorders) | 0 (0) | 1 (1)
Dysaesthesia (Nervous system disorders) | 14 (15) | 7 (8)
Dysarthria (Nervous system disorders) | 1 (2) | 1 (1)
Dysgeusia (Nervous system disorders) | 72 (81) | 14 (14)
Dysgraphia (Nervous system disorders) | 1 (1) | 0 (0)
Dyskinesia (Nervous system disorders) | 2 (2) | 4 (4)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 1 (1)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Facial neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 1 (1) | 2 (2)
Head discomfort (Nervous system disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 445 (590) | 338 (405)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 8 (8) | 3 (3)
Hypersomnia (Nervous system disorders) | 4 (4) | 1 (1)
Hypertonia (Nervous system disorders) | 1 (1) | 3 (3)
Hypoaesthesia (Nervous system disorders) | 30 (38) | 31 (35)
Hypokinesia (Nervous system disorders) | 1 (1) | 0 (0)
Hyposmia (Nervous system disorders) | 2 (2) | 1 (1)
Intercostal neuralgia (Nervous system disorders) | 3 (3) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 14 (16) | 7 (7)
Memory impairment (Nervous system disorders) | 46 (50) | 59 (64)
Mental impairment (Nervous system disorders) | 1 (1) | 1 (1)
Migraine (Nervous system disorders) | 27 (32) | 21 (23)
Migraine with aura (Nervous system disorders) | 2 (2) | 0 (0)
Morton's neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Muscle contractions involuntary (Nervous system disorders) | 2 (3) | 0 (0)
Muscle spasticity (Nervous system disorders) | 2 (2) | 1 (1)
Myoclonus (Nervous system disorders) | 0 (0) | 1 (1)
Nerve compression (Nervous system disorders) | 0 (0) | 3 (4)
Nervous system disorder (Nervous system disorders) | 1 (1) | 1 (2)
Neuralgia (Nervous system disorders) | 21 (21) | 15 (15)
Neuritis (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 148 (186) | 102 (121)
Neurotoxicity (Nervous system disorders) | 10 (10) | 11 (11)
Occipital neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 115 (129) | 82 (89)
Paresis (Nervous system disorders) | 1 (1) | 0 (0)
Parkinson's disease (Nervous system disorders) | 1 (1) | 2 (2)
Parosmia (Nervous system disorders) | 1 (1) | 0 (0)
Partial seizures (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 8 (11) | 7 (7)
Peripheral nerve lesion (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 65 (78) | 49 (53)
Petit mal epilepsy (Nervous system disorders) | 1 (1) | 1 (1)
Phantom limb syndrome (Nervous system disorders) | 2 (2) | 0 (0)
Polyneuropathy (Nervous system disorders) | 12 (14) | 12 (14)
Poor quality sleep (Nervous system disorders) | 2 (2) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 2 (3) | 1 (1)
Presyncope (Nervous system disorders) | 9 (9) | 3 (3)
Radicular pain (Nervous system disorders) | 1 (1) | 0 (0)
Resting tremor (Nervous system disorders) | 1 (1) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 7 (7) | 9 (9)
Sciatica (Nervous system disorders) | 19 (20) | 19 (22)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Sensorimotor disorder (Nervous system disorders) | 1 (1) | 0 (0)
Sensory disturbance (Nervous system disorders) | 2 (2) | 0 (0)
Sinus headache (Nervous system disorders) | 6 (7) | 4 (4)
Somnolence (Nervous system disorders) | 7 (7) | 7 (7)
Speech disorder (Nervous system disorders) | 0 (0) | 1 (1)
Spinal cord herniation (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 23 (23) | 17 (19)
Taste disorder (Nervous system disorders) | 27 (29) | 4 (4)
Tension headache (Nervous system disorders) | 4 (4) | 3 (3)
Thoracic outlet syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 14 (14) | 12 (13)
Trigeminal neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Visual field defect (Nervous system disorders) | 1 (1) | 0 (0)
Device failure (Product Issues) | 1 (1) | 0 (0)
Device leakage (Product Issues) | 0 (0) | 1 (1)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 2 (2)
Adjustment disorder with depressed mood (Psychiatric disorders) | 2 (2) | 1 (1)
Adjustment disorder with mixed disturbance of emotion and conduct (Psychiatric disorders) | 0 (0) | 1 (1)
Affect lability (Psychiatric disorders) | 9 (10) | 17 (20)
Affective disorder (Psychiatric disorders) | 0 (0) | 3 (3)
Aggression (Psychiatric disorders) | 1 (1) | 0 (0)
Agitated depression (Psychiatric disorders) | 1 (1) | 1 (1)
Agitation (Psychiatric disorders) | 22 (22) | 12 (12)
Agoraphobia (Psychiatric disorders) | 1 (1) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 2 (3) | 0 (0)
Anger (Psychiatric disorders) | 0 (0) | 1 (1)
Anhedonia (Psychiatric disorders) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 157 (184) | 143 (168)
Anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Apathy (Psychiatric disorders) | 1 (1) | 0 (0)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 1 (1) | 3 (3)
Bradyphrenia (Psychiatric disorders) | 1 (1) | 4 (4)
Bruxism (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 7 (7) | 5 (6)
Conversion disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Daydreaming (Psychiatric disorders) | 1 (1) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 38 (44) | 33 (39)
Depression (Psychiatric disorders) | 156 (191) | 150 (175)
Depressive symptom (Psychiatric disorders) | 0 (0) | 2 (2)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1)
Eating disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Emotional disorder (Psychiatric disorders) | 0 (0) | 2 (2)
Emotional distress (Psychiatric disorders) | 1 (1) | 3 (3)
Female orgasmic disorder (Psychiatric disorders) | 0 (0) | 1 (2)
Flashback (Psychiatric disorders) | 0 (0) | 1 (1)
Genito-pelvic pain/penetration disorder (Psychiatric disorders) | 2 (2) | 0 (0)
Hallucination, auditory (Psychiatric disorders) | 0 (0) | 1 (1)
Initial insomnia (Psychiatric disorders) | 2 (3) | 2 (2)
Insomnia (Psychiatric disorders) | 383 (468) | 357 (418)
Irritability (Psychiatric disorders) | 30 (34) | 25 (28)
Libido decreased (Psychiatric disorders) | 31 (33) | 34 (38)
Libido disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Loss of libido (Psychiatric disorders) | 1 (1) | 2 (2)
Mania (Psychiatric disorders) | 1 (1) | 0 (0)
Mental disorder (Psychiatric disorders) | 3 (3) | 0 (0)
Middle insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Mixed anxiety and depressive disorder (Psychiatric disorders) | 2 (2) | 5 (5)
Mood altered (Psychiatric disorders) | 20 (23) | 26 (28)
Mood swings (Psychiatric disorders) | 20 (24) | 28 (30)
Negative thoughts (Psychiatric disorders) | 1 (1) | 0 (0)
Nervousness (Psychiatric disorders) | 3 (3) | 3 (3)
Nightmare (Psychiatric disorders) | 2 (3) | 1 (1)
Orgasm abnormal (Psychiatric disorders) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 5 (5) | 3 (3)
Paranoia (Psychiatric disorders) | 0 (0) | 1 (1)
Perinatal depression (Psychiatric disorders) | 0 (0) | 1 (1)
Persistent depressive disorder (Psychiatric disorders) | 4 (5) | 1 (2)
Personality change (Psychiatric disorders) | 2 (2) | 0 (0)
Phonophobia (Psychiatric disorders) | 0 (0) | 1 (1)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 3 (3)
Seasonal affective disorder (Psychiatric disorders) | 0 (0) | 2 (2)
Sleep disorder (Psychiatric disorders) | 24 (31) | 26 (33)
Stress (Psychiatric disorders) | 1 (1) | 7 (7)
Suicidal ideation (Psychiatric disorders) | 2 (2) | 4 (4)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Tearfulness (Psychiatric disorders) | 2 (3) | 1 (1)
Terminal insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Thinking abnormal (Psychiatric disorders) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 4 (5)
Bladder discomfort (Renal and urinary disorders) | 1 (1) | 1 (1)
Bladder dysfunction (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder prolapse (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 2 (2) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1)
Chromaturia (Renal and urinary disorders) | 2 (2) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 4 (7) | 9 (10)
Cystitis noninfective (Renal and urinary disorders) | 3 (3) | 1 (1)
Dysuria (Renal and urinary disorders) | 36 (43) | 18 (21)
Haematuria (Renal and urinary disorders) | 13 (13) | 12 (13)
Hydronephrosis (Renal and urinary disorders) | 2 (2) | 0 (0)
Hypercalciuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Hypertonic bladder (Renal and urinary disorders) | 1 (1) | 2 (2)
Incontinence (Renal and urinary disorders) | 2 (2) | 2 (2)
Leukocyturia (Renal and urinary disorders) | 1 (1) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 7 (7) | 8 (10)
Nephrolithiasis (Renal and urinary disorders) | 6 (6) | 9 (10)
Nocturia (Renal and urinary disorders) | 6 (6) | 3 (3)
Pollakiuria (Renal and urinary disorders) | 30 (33) | 21 (23)
Polyuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1) | 4 (4)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 3 (3) | 0 (0)
Renal injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal mass (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal pain (Renal and urinary disorders) | 2 (2) | 2 (2)
Strangury (Renal and urinary disorders) | 0 (0) | 1 (1)
Stress urinary incontinence (Renal and urinary disorders) | 3 (3) | 2 (2)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureteric stenosis (Renal and urinary disorders) | 1 (4) | 0 (0)
Urge incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary bladder polyp (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary hesitation (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 19 (22) | 22 (27)
Urinary retention (Renal and urinary disorders) | 1 (1) | 2 (2)
Urinary tract disorder (Renal and urinary disorders) | 1 (1) | 2 (2)
Urinary tract inflammation (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary tract pain (Renal and urinary disorders) | 9 (9) | 7 (9)
Urine flow decreased (Renal and urinary disorders) | 1 (1) | 0 (0)
Urine odour abnormal (Renal and urinary disorders) | 3 (3) | 0 (0)
Adnexa uteri pain (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Amenorrhoea (Reproductive system and breast disorders) | 2 (2) | 3 (3)
Anisomastia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 6 (9) | 11 (11)
Bartholin's cyst (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Breast calcifications (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Breast cyst (Reproductive system and breast disorders) | 3 (3) | 3 (3)
Breast discharge (Reproductive system and breast disorders) | 3 (4) | 1 (1)
Breast discomfort (Reproductive system and breast disorders) | 15 (16) | 9 (9)
Breast disorder (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Breast fibrosis (Reproductive system and breast disorders) | 5 (5) | 10 (10)
Breast haematoma (Reproductive system and breast disorders) | 5 (5) | 3 (3)
Breast hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast induration (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Breast inflammation (Reproductive system and breast disorders) | 2 (2) | 3 (3)
Breast mass (Reproductive system and breast disorders) | 12 (13) | 10 (10)
Breast necrosis (Reproductive system and breast disorders) | 4 (4) | 1 (1)
Breast oedema (Reproductive system and breast disorders) | 20 (21) | 18 (18)
Breast pain (Reproductive system and breast disorders) | 145 (163) | 158 (186)
Breast swelling (Reproductive system and breast disorders) | 7 (7) | 13 (14)
Breast tenderness (Reproductive system and breast disorders) | 2 (2) | 17 (17)
Breast ulceration (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Cervical polyp (Reproductive system and breast disorders) | 3 (3) | 1 (1)
Coital bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 3 (3) | 4 (4)
Dyspareunia (Reproductive system and breast disorders) | 37 (43) | 35 (38)
Endometrial atrophy (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Endometrial disorder (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Endometrial hyperplasia (Reproductive system and breast disorders) | 8 (8) | 9 (9)
Endometrial hypertrophy (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Endometrial thickening (Reproductive system and breast disorders) | 2 (3) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Fibrocystic breast disease (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Genital haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Genital lesion (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Menopausal disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Menopausal symptoms (Reproductive system and breast disorders) | 6 (7) | 2 (2)
Menorrhagia (Reproductive system and breast disorders) | 7 (7) | 12 (15)
Menstrual disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 7 (7) | 9 (10)
Metrorrhagia (Reproductive system and breast disorders) | 3 (3) | 5 (5)
Nipple disorder (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Nipple exudate bloody (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Nipple pain (Reproductive system and breast disorders) | 0 (0) | 4 (4)
Ovarian cyst (Reproductive system and breast disorders) | 7 (7) | 12 (13)
Ovarian disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic adhesions (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic floor muscle weakness (Reproductive system and breast disorders) | 1 (1) | 4 (4)
Pelvic pain (Reproductive system and breast disorders) | 16 (18) | 21 (23)
Perineal pain (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Premature menopause (Reproductive system and breast disorders) | 1 (1) | 3 (3)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Reproductive tract disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Retracted nipple (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Uterine haemorrhage (Reproductive system and breast disorders) | 1 (1) | 1 (2)
Uterine polyp (Reproductive system and breast disorders) | 5 (5) | 7 (8)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine spasm (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 31 (32) | 42 (49)
Vaginal haemorrhage (Reproductive system and breast disorders) | 43 (46) | 68 (79)
Vaginal lesion (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal prolapse (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 3 (3) | 1 (1)
Vulvovaginal dryness (Reproductive system and breast disorders) | 182 (211) | 213 (254)
Vulvovaginal inflammation (Reproductive system and breast disorders) | 1 (1) | 3 (3)
Vulvovaginal pain (Reproductive system and breast disorders) | 3 (3) | 4 (5)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 12 (15) | 11 (14)
Allergic bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Allergic respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Aphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 4 (4)
Asthma exercise induced (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Bronchial disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (3)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 5 (6)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 416 (543) | 222 (256)
Cough variant asthma (Respiratory, thoracic and mediastinal disorders) | 1 (5) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 29 (31) | 9 (9)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 197 (247) | 130 (144)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 31 (31) | 12 (12)
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 108 (131) | 16 (16)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 0 (0)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 2 (2)
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Lymphangioleiomyomatosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 98 (118) | 26 (29)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 0 (0)
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 18 (19) | 1 (1)
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal pruritus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 155 (169) | 60 (65)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal paraesthesia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 3 (3)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 5 (5)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 41 (45) | 21 (24)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 4 (4)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Respiratory tract irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 42 (48) | 24 (25)
Rhinitis atrophic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 52 (56) | 16 (16)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 4 (4)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 4 (4)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 5 (9) | 9 (9)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1)
Throat lesion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (5)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tonsillar ulcer (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tonsillolith (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Upper respiratory tract irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 32 (36) | 19 (20)
Vocal cord atrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vocal cord dysfunction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 7 (10) | 10 (15)
Acne (Skin and subcutaneous tissue disorders) | 11 (12) | 4 (5)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 510 (558) | 149 (163)
Alopecia totalis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 11 (13) | 2 (2)
Blood blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Capillaritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Chloasma (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Chronic pigmented purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Cold sweat (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Cutaneous symptom (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 4 (4) | 7 (7)
Dermatitis (Skin and subcutaneous tissue disorders) | 11 (11) | 12 (12)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 32 (39) | 13 (15)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Dermatomyositis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (5) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 153 (178) | 56 (67)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 22 (24) | 13 (14)
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 54 (56) | 42 (45)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3 (5) | 1 (1)
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hirsutism (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 38 (40) | 31 (36)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)
Hypertrophic scar (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Idiopathic urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (3)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Itching scar (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Keloid scar (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Lichen planus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3)
Lichen sclerosus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Madarosis (Skin and subcutaneous tissue disorders) | 22 (25) | 4 (4)
Milia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Miliaria (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Myxoid cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Nail bed disorder (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Nail bed inflammation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail discolouration (Skin and subcutaneous tissue disorders) | 9 (9) | 3 (3)
Nail disorder (Skin and subcutaneous tissue disorders) | 31 (35) | 11 (13)
Nail dystrophy (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Nail ridging (Skin and subcutaneous tissue disorders) | 10 (10) | 3 (3)
Nail toxicity (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Night sweats (Skin and subcutaneous tissue disorders) | 42 (50) | 50 (53)
Onychalgia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Onychoclasis (Skin and subcutaneous tissue disorders) | 29 (29) | 3 (3)
Onycholysis (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3)
Onychomadesis (Skin and subcutaneous tissue disorders) | 16 (16) | 9 (9)
Pain of skin (Skin and subcutaneous tissue disorders) | 14 (15) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 10 (11) | 1 (1)
Panniculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Papule (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Papulopustular rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Peau d'orange (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (1)
Photodermatosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 7 (7) | 2 (2)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Plantar erythema (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Prurigo (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 183 (222) | 95 (105)
Psoriasis (Skin and subcutaneous tissue disorders) | 7 (10) | 7 (7)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 229 (288) | 90 (102)
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (5)
Rash follicular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 6 (6) | 3 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 65 (108) | 25 (32)
Rash papular (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 12 (12) | 9 (11)
Rosacea (Skin and subcutaneous tissue disorders) | 10 (10) | 4 (4)
Scab (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Scar pain (Skin and subcutaneous tissue disorders) | 15 (16) | 23 (26)
Sebaceous hyperplasia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Sensitive skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin atrophy (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Skin discolouration (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (4)
Skin discomfort (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 4 (5) | 9 (10)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 10 (10) | 4 (4)
Skin fissures (Skin and subcutaneous tissue disorders) | 7 (8) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 11 (13) | 17 (18)
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Skin induration (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Skin irritation (Skin and subcutaneous tissue disorders) | 7 (7) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 17 (18) | 9 (11)
Skin mass (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Skin oedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin plaque (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin striae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin tightness (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Skin toxicity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 7 (9) | 2 (2)
Skin warm (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin weeping (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Solar lentigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Trichorrhexis (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 24 (29) | 11 (12)
Vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Xeroderma (Skin and subcutaneous tissue disorders) | 2 (5) | 2 (2)
Postmenopause (Social circumstances) | 1 (1) | 0 (0)
Sight disability (Social circumstances) | 2 (2) | 0 (0)
Breast operation (Surgical and medical procedures) | 3 (3) | 1 (1)
Breast prosthesis removal (Surgical and medical procedures) | 1 (1) | 1 (1)
Breast reconstruction (Surgical and medical procedures) | 9 (11) | 7 (9)
Cataract operation (Surgical and medical procedures) | 1 (1) | 2 (2)
Central venous catheter removal (Surgical and medical procedures) | 1 (1) | 2 (2)
Cholecystectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Dental care (Surgical and medical procedures) | 1 (2) | 0 (0)
Dental operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Drain removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Endodontic procedure (Surgical and medical procedures) | 0 (0) | 1 (1)
Hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Hysterosalpingo-oophorectomy (Surgical and medical procedures) | 1 (1) | 1 (1)
Incisional drainage (Surgical and medical procedures) | 2 (2) | 1 (1)
Infection prophylaxis (Surgical and medical procedures) | 1 (1) | 0 (0)
Joint dislocation reduction (Surgical and medical procedures) | 0 (0) | 1 (1)
Lipoma excision (Surgical and medical procedures) | 1 (1) | 0 (0)
Mammoplasty (Surgical and medical procedures) | 2 (2) | 0 (0)
Medical device removal (Surgical and medical procedures) | 0 (0) | 1 (1)
Medical procedure (Surgical and medical procedures) | 1 (1) | 0 (0)
Meniscus operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Metabolic surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Micrographic skin surgery (Surgical and medical procedures) | 1 (2) | 0 (0)
Mole excision (Surgical and medical procedures) | 2 (2) | 1 (1)
Nail operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Oophorectomy (Surgical and medical procedures) | 2 (2) | 0 (0)
Post procedural drainage (Surgical and medical procedures) | 1 (1) | 1 (2)
Salpingo-oophorectomy bilateral (Surgical and medical procedures) | 1 (1) | 2 (2)
Sinus operation (Surgical and medical procedures) | 5 (5) | 0 (0)
Skin lesion removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Skin neoplasm excision (Surgical and medical procedures) | 1 (1) | 0 (0)
Spinal operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgery (Surgical and medical procedures) | 4 (5) | 1 (1)
Tendon sheath incision (Surgical and medical procedures) | 0 (0) | 1 (1)
Thyroid operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 2 (3) | 0 (0)
Weight loss diet (Surgical and medical procedures) | 3 (3) | 1 (1)
Wound drainage (Surgical and medical procedures) | 3 (3) | 0 (0)
Angiopathy (Vascular disorders) | 2 (2) | 3 (3)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Aortic arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Aortic dilatation (Vascular disorders) | 1 (1) | 1 (1)
Arterial thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Arteriovenous fistula (Vascular disorders) | 0 (0) | 1 (1)
Axillary vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Bleeding varicose vein (Vascular disorders) | 0 (0) | 1 (1)
Blood pressure inadequately controlled (Vascular disorders) | 0 (0) | 1 (1)
Capillary fragility (Vascular disorders) | 5 (5) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 9 (9) | 5 (8)
Embolism (Vascular disorders) | 9 (9) | 3 (4)
Essential hypertension (Vascular disorders) | 0 (0) | 1 (2)
Flushing (Vascular disorders) | 15 (20) | 24 (33)
Haematoma (Vascular disorders) | 20 (20) | 7 (7)
Hot flush (Vascular disorders) | 702 (887) | 849 (1066)
Hypertension (Vascular disorders) | 205 (363) | 227 (382)
Hypertensive crisis (Vascular disorders) | 2 (3) | 1 (1)
Hypotension (Vascular disorders) | 28 (31) | 16 (16)
Intermittent claudication (Vascular disorders) | 1 (1) | 0 (0)
Lymphocele (Vascular disorders) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 336 (395) | 268 (303)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 2 (2)
Peripheral coldness (Vascular disorders) | 3 (3) | 3 (3)
Peripheral venous disease (Vascular disorders) | 6 (7) | 2 (2)
Phlebitis (Vascular disorders) | 6 (7) | 6 (8)
Poor peripheral circulation (Vascular disorders) | 2 (2) | 0 (0)
Post thrombotic syndrome (Vascular disorders) | 1 (1) | 0 (0)
Prehypertension (Vascular disorders) | 0 (0) | 1 (1)
Raynaud's phenomenon (Vascular disorders) | 3 (4) | 1 (1)
Subclavian vein thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Thrombophlebitis (Vascular disorders) | 5 (7) | 3 (3)
Thrombophlebitis superficial (Vascular disorders) | 5 (6) | 5 (5)
Thrombosis (Vascular disorders) | 8 (11) | 2 (2)
Varicophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Varicose vein (Vascular disorders) | 4 (4) | 4 (5)
Venous thrombosis (Vascular disorders) | 1 (2) | 0 (0)
White coat hypertension (Vascular disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-23): https://cdn.clinicaltrials.gov/large-docs/94/NCT02513394/Prot_SAP_000.pdf